CLINICAL TRIAL: NCT04922216
Title: Optimization of a mHealth Behavioral Weight Loss Intervention for Young Adults
Brief Title: Adaptive Goals and Interventions for Lifestyle Enhancement
Acronym: AGILE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 20-0765; R01DK125779 (NIH)
Record Dates: First submitted 2021-06-04; First posted 2021-06-10 (Actual); Results first posted 2025-07-20 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2023-10

CONDITIONS: Obesity
Keywords: behavioral intervention; JITAI (just-in-time adaptive intervention)
MeSH Terms: conditions — Obesity | interventions — YES1 protein, human

STUDY DESIGN:
Intervention Model Description: This study uses a full factorial experimental design testing the efficacy of five intervention components, each with two levels
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (32):
- Condition 1 (Experimental): Core + Standard Diet Monitoring + Daily Activity Goal + Fixed Timing + Standard Content + No Choice
  Interventions: Behavioral: Core; Behavioral: Standard Diet Monitoring; Behavioral: Adaptive Activity Goals (Daily); Behavioral: Message Decision Points (Fixed); Behavioral: Message Decision Rules (Standard); Behavioral: Message Choice (No)
- Condition 2 (Experimental): Core + Standard Diet Monitoring + Daily Activity Goal + Fixed Timing + Standard Content + Choice
  Interventions: Behavioral: Core; Behavioral: Standard Diet Monitoring; Behavioral: Adaptive Activity Goals (Daily); Behavioral: Message Decision Points (Fixed); Behavioral: Message Decision Rules (Standard); Behavioral: Message Choice (Yes)
- Condition 3 (Experimental): Core + Standard Diet Monitoring + Daily Activity Goal + Fixed Timing + Adaptive Content + No Choice
  Interventions: Behavioral: Core; Behavioral: Standard Diet Monitoring; Behavioral: Adaptive Activity Goals (Daily); Behavioral: Message Decision Points (Fixed); Behavioral: Message Decision Rules (Adaptive); Behavioral: Message Choice (No)
- Condition 4 (Experimental): Core + Standard Diet Monitoring + Daily Activity Goal + Fixed Timing + Adaptive Content + Choice
  Interventions: Behavioral: Core; Behavioral: Standard Diet Monitoring; Behavioral: Adaptive Activity Goals (Daily); Behavioral: Message Decision Points (Fixed); Behavioral: Message Decision Rules (Adaptive); Behavioral: Message Choice (Yes)
- Condition 5 (Experimental): Core+Standard Diet Monitoring+Daily Activity Goal+Adaptive Timing+Standard Content+No Choice
  Interventions: Behavioral: Core; Behavioral: Standard Diet Monitoring; Behavioral: Adaptive Activity Goals (Daily); Behavioral: Message Decision Points (Adaptive); Behavioral: Message Decision Rules (Standard); Behavioral: Message Choice (No)
- Condition 6 (Experimental): Core + Standard Diet Monitoring + Daily Activity Goal + Adaptive Timing + Standard Content + Choice
  Interventions: Behavioral: Core; Behavioral: Standard Diet Monitoring; Behavioral: Adaptive Activity Goals (Daily); Behavioral: Message Decision Points (Adaptive); Behavioral: Message Decision Rules (Standard); Behavioral: Message Choice (Yes)
- Condition 7 (Experimental): Core+ Standard Diet Monitoring+ Daily Activity Goal+ Adaptive Timing+ Adaptive Content+ No Choice
  Interventions: Behavioral: Core; Behavioral: Standard Diet Monitoring; Behavioral: Adaptive Activity Goals (Daily); Behavioral: Message Decision Points (Adaptive); Behavioral: Message Decision Rules (Adaptive); Behavioral: Message Choice (No)
- Condition 8 (Experimental): Core + Standard Diet Monitoring + Daily Activity Goal + Adaptive Timing + Adaptive Content + Choice
  Interventions: Behavioral: Core; Behavioral: Standard Diet Monitoring; Behavioral: Adaptive Activity Goals (Daily); Behavioral: Message Decision Points (Adaptive); Behavioral: Message Decision Rules (Adaptive); Behavioral: Message Choice (Yes)
- Condition 9 (Experimental): Core + Standard Diet Monitoring + Weekly Activity Goal + Fixed Timing + Standard Content + No Choice
  Interventions: Behavioral: Core; Behavioral: Standard Diet Monitoring; Behavioral: Adaptive Activity Goals (Weekly); Behavioral: Message Decision Points (Fixed); Behavioral: Message Decision Rules (Standard); Behavioral: Message Choice (No)
- Condition 10 (Experimental): Core + Standard Diet Monitoring + Weekly Activity Goal + Fixed Timing + Standard Content + Choice
  Interventions: Behavioral: Core; Behavioral: Standard Diet Monitoring; Behavioral: Adaptive Activity Goals (Weekly); Behavioral: Message Decision Points (Fixed); Behavioral: Message Decision Rules (Standard); Behavioral: Message Choice (Yes)
- Condition 11 (Experimental): Core + Standard Diet Monitoring + Weekly Activity Goal + Fixed Timing + Adaptive Content + No Choice
  Interventions: Behavioral: Core; Behavioral: Standard Diet Monitoring; Behavioral: Adaptive Activity Goals (Weekly); Behavioral: Message Decision Points (Fixed); Behavioral: Message Decision Rules (Adaptive); Behavioral: Message Choice (No)
- Condition 12 (Experimental): Core + Standard Diet Monitoring + Weekly Activity Goal + Fixed Timing + Adaptive Content + Choice
  Interventions: Behavioral: Core; Behavioral: Standard Diet Monitoring; Behavioral: Adaptive Activity Goals (Weekly); Behavioral: Message Decision Points (Fixed); Behavioral: Message Decision Rules (Adaptive); Behavioral: Message Choice (Yes)
- Condition 13 (Experimental): Core+Standard Diet Monitoring+Weekly Activity Goal+Adaptive Timing+Standard Content+No Choice
  Interventions: Behavioral: Core; Behavioral: Standard Diet Monitoring; Behavioral: Adaptive Activity Goals (Weekly); Behavioral: Message Decision Points (Adaptive); Behavioral: Message Decision Rules (Standard); Behavioral: Message Choice (No)
- Condition 14 (Experimental): Core + Standard Diet Monitoring + Weekly Activity Goal + Adaptive Timing + Standard Content + Choice
  Interventions: Behavioral: Core; Behavioral: Standard Diet Monitoring; Behavioral: Adaptive Activity Goals (Weekly); Behavioral: Message Decision Points (Adaptive); Behavioral: Message Decision Rules (Standard); Behavioral: Message Choice (Yes)
- Condition 15 (Experimental): Core + Standard Diet Monitoring+ Weekly Activity Goal+ Adaptive Timing+ Adaptive Content+ No Choice
  Interventions: Behavioral: Core; Behavioral: Standard Diet Monitoring; Behavioral: Adaptive Activity Goals (Weekly); Behavioral: Message Decision Points (Adaptive); Behavioral: Message Decision Rules (Adaptive); Behavioral: Message Choice (No)
- Condition 16 (Experimental): Core + Standard Diet Monitoring + Weekly Activity Goal + Adaptive Timing + Adaptive Content + Choice
  Interventions: Behavioral: Core; Behavioral: Standard Diet Monitoring; Behavioral: Adaptive Activity Goals (Weekly); Behavioral: Message Decision Points (Adaptive); Behavioral: Message Decision Rules (Adaptive); Behavioral: Message Choice (Yes)
- Condition 17 (Experimental): Core+ Simplified Diet Monitoring+ Daily Activity Goal+ Fixed Timing+ Standard Content+ No Choice
  Interventions: Behavioral: Core; Behavioral: Simplified Diet Monitoring; Behavioral: Adaptive Activity Goals (Daily); Behavioral: Message Decision Points (Fixed); Behavioral: Message Decision Rules (Standard); Behavioral: Message Choice (No)
- Condition 18 (Experimental): Core+ Simplified Diet Monitoring+ Daily Activity Goal+ Fixed Timing+ Standard Content+ Choice
  Interventions: Behavioral: Core; Behavioral: Simplified Diet Monitoring; Behavioral: Adaptive Activity Goals (Daily); Behavioral: Message Decision Points (Fixed); Behavioral: Message Decision Rules (Standard); Behavioral: Message Choice (Yes)
- Condition 19 (Experimental): Core+ Simplified Diet Monitoring+ Daily Activity Goal+ Fixed Timing+ Adaptive Content+ No Choice
  Interventions: Behavioral: Core; Behavioral: Simplified Diet Monitoring; Behavioral: Adaptive Activity Goals (Daily); Behavioral: Message Decision Points (Fixed); Behavioral: Message Decision Rules (Adaptive); Behavioral: Message Choice (No)
- Condition 20 (Experimental): Core + Simplified Diet Monitoring + Daily Activity Goal + Fixed Timing + Adaptive Content + Choice
  Interventions: Behavioral: Core; Behavioral: Simplified Diet Monitoring; Behavioral: Adaptive Activity Goals (Daily); Behavioral: Message Decision Points (Fixed); Behavioral: Message Decision Rules (Adaptive); Behavioral: Message Choice (Yes)
- Condition 21 (Experimental): Core+ Simplified Diet Monitoring+ Daily Activity Goal+ Adaptive Timing+ Standard Content+ No Choice
  Interventions: Behavioral: Core; Behavioral: Simplified Diet Monitoring; Behavioral: Adaptive Activity Goals (Daily); Behavioral: Message Decision Points (Adaptive); Behavioral: Message Decision Rules (Standard); Behavioral: Message Choice (No)
- Condition 22 (Experimental): Core+ Simplified Diet Monitoring+ Daily Activity Goal+ Adaptive Timing+ Standard Content+ Choice
  Interventions: Behavioral: Core; Behavioral: Simplified Diet Monitoring; Behavioral: Adaptive Activity Goals (Daily); Behavioral: Message Decision Points (Adaptive); Behavioral: Message Decision Rules (Standard); Behavioral: Message Choice (Yes)
- Condition 23 (Experimental): Core+ Simplified Diet Monitoring+ Daily Activity Goal+ Adaptive Timing+ Adaptive Content+ No Choice
  Interventions: Behavioral: Core; Behavioral: Simplified Diet Monitoring; Behavioral: Adaptive Activity Goals (Daily); Behavioral: Message Decision Points (Adaptive); Behavioral: Message Decision Rules (Adaptive); Behavioral: Message Choice (No)
- Condition 24 (Experimental): Core+ Simplified Diet Monitoring+ Daily Activity Goal+ Adaptive Timing+ Adaptive Content+ Choice
  Interventions: Behavioral: Core; Behavioral: Simplified Diet Monitoring; Behavioral: Adaptive Activity Goals (Daily); Behavioral: Message Decision Points (Adaptive); Behavioral: Message Decision Rules (Adaptive); Behavioral: Message Choice (Yes)
- Condition 25 (Experimental): Core+ Simplified Diet Monitoring+ Weekly Activity Goal+ Fixed Timing+ Standard Content+ No Choice
  Interventions: Behavioral: Core; Behavioral: Simplified Diet Monitoring; Behavioral: Adaptive Activity Goals (Weekly); Behavioral: Message Decision Points (Fixed); Behavioral: Message Decision Rules (Standard); Behavioral: Message Choice (No)
- Condition 26 (Experimental): Core + Simplified Diet Monitoring + Weekly Activity Goal + Fixed Timing + Standard Content + Choice
  Interventions: Behavioral: Core; Behavioral: Simplified Diet Monitoring; Behavioral: Adaptive Activity Goals (Weekly); Behavioral: Message Decision Points (Fixed); Behavioral: Message Decision Rules (Standard); Behavioral: Message Choice (Yes)
- Condition 27 (Experimental): Core+ Simplified Diet Monitoring+ Weekly Activity Goal+ Fixed Timing+ Adaptive Content+ No Choice
  Interventions: Behavioral: Core; Behavioral: Simplified Diet Monitoring; Behavioral: Adaptive Activity Goals (Weekly); Behavioral: Message Decision Points (Fixed); Behavioral: Message Decision Rules (Adaptive); Behavioral: Message Choice (No)
- Condition 28 (Experimental): Core + Simplified Diet Monitoring + Weekly Activity Goal + Fixed Timing + Adaptive Content + Choice
  Interventions: Behavioral: Core; Behavioral: Simplified Diet Monitoring; Behavioral: Adaptive Activity Goals (Weekly); Behavioral: Message Decision Points (Fixed); Behavioral: Message Decision Rules (Adaptive); Behavioral: Message Choice (Yes)
- Condition 29 (Experimental): Core+ Simplified Diet Monitoring+ Weekly Activity Goal+ Adaptive Timing+ Standard Content+ No Choice
  Interventions: Behavioral: Core; Behavioral: Simplified Diet Monitoring; Behavioral: Adaptive Activity Goals (Weekly); Behavioral: Message Decision Points (Adaptive); Behavioral: Message Decision Rules (Standard); Behavioral: Message Choice (No)
- Condition 30 (Experimental): Core+ Simplified Diet Monitoring+ Weekly Activity Goal+ Adaptive Timing+ Standard Content+ Choice
  Interventions: Behavioral: Core; Behavioral: Simplified Diet Monitoring; Behavioral: Adaptive Activity Goals (Weekly); Behavioral: Message Decision Points (Adaptive); Behavioral: Message Decision Rules (Standard); Behavioral: Message Choice (Yes)
- Condition 31 (Experimental): Core+ Simplified Diet Monitoring+ Weekly Activity Goal+ Adaptive Timing+ Adaptive Content+ No Choice
  Interventions: Behavioral: Core; Behavioral: Simplified Diet Monitoring; Behavioral: Adaptive Activity Goals (Weekly); Behavioral: Message Decision Points (Adaptive); Behavioral: Message Decision Rules (Adaptive); Behavioral: Message Choice (No)
- Condition 32 (Experimental): Core + Simplified Diet Monitoring + Weekly Activity Goal + Adaptive Timing + Adaptive Content+Choice
  Interventions: Behavioral: Core; Behavioral: Simplified Diet Monitoring; Behavioral: Adaptive Activity Goals (Weekly); Behavioral: Message Decision Points (Adaptive); Behavioral: Message Decision Rules (Adaptive); Behavioral: Message Choice (Yes)

INTERVENTIONS:
Behavioral: Core — Behavioral weight loss core includes behavioral lessons, activity tracker, daily self-weighing, weekly tailored feedback summary.
Behavioral: Standard Diet Monitoring — Standard monitoring using smartphone tracking of all calorie intake.
  Arms: Condition 1; Condition 10; Condition 11; Condition 12; Condition 13; Condition 14; Condition 15; Condition 16; Condition 2; Condition 3; Condition 4; Condition 5; Condition 6; Condition 7; Condition 8; Condition 9
Behavioral: Simplified Diet Monitoring — Simplified diet monitoring using smartphone tracking of red foods using a traffic light approach.
  Arms: Condition 17; Condition 18; Condition 19; Condition 20; Condition 21; Condition 22; Condition 23; Condition 24; Condition 25; Condition 26; Condition 27; Condition 28; Condition 29; Condition 30; Condition 31; Condition 32
Behavioral: Adaptive Activity Goals (Daily) — Physical activity goals that adapt once each day using the participants' data derived from activity tracker.
  Arms: Condition 1; Condition 17; Condition 18; Condition 19; Condition 2; Condition 20; Condition 21; Condition 22; Condition 23; Condition 24; Condition 3; Condition 4; Condition 5; Condition 6; Condition 7; Condition 8
Behavioral: Adaptive Activity Goals (Weekly) — Physical activity goals that adapt once each week using the participants' data derived from activity tracker.
  Arms: Condition 10; Condition 11; Condition 12; Condition 13; Condition 14; Condition 15; Condition 16; Condition 25; Condition 26; Condition 27; Condition 28; Condition 29; Condition 30; Condition 31; Condition 32; Condition 9
Behavioral: Message Decision Points (Fixed) — Message timing is fixed and evaluated at specific times each day to determine message eligibility.
  Arms: Condition 1; Condition 10; Condition 11; Condition 12; Condition 17; Condition 18; Condition 19; Condition 2; Condition 20; Condition 25; Condition 26; Condition 27; Condition 28; Condition 3; Condition 4; Condition 9
Behavioral: Message Decision Points (Adaptive) — Message timing is adaptive and derived from individual user data to determine message eligibility.
  Arms: Condition 13; Condition 14; Condition 15; Condition 16; Condition 21; Condition 22; Condition 23; Condition 24; Condition 29; Condition 30; Condition 31; Condition 32; Condition 5; Condition 6; Condition 7; Condition 8
Behavioral: Message Decision Rules (Standard) — Decision rules to determine eligibility to receive just-in-time messages consider participant's recent behaviors.
  Arms: Condition 1; Condition 10; Condition 13; Condition 14; Condition 17; Condition 18; Condition 2; Condition 21; Condition 22; Condition 25; Condition 26; Condition 29; Condition 30; Condition 5; Condition 6; Condition 9
Behavioral: Message Decision Rules (Adaptive) — Decision rules to determine eligibility to receive just-in-time messages consider participant's recent behaviors and overall progress.
  Arms: Condition 11; Condition 12; Condition 15; Condition 16; Condition 19; Condition 20; Condition 23; Condition 24; Condition 27; Condition 28; Condition 3; Condition 31; Condition 32; Condition 4; Condition 7; Condition 8
Behavioral: Message Choice (No) — Participant choice does not drive adaptation of 1) message type delivered or 2) lapse support provision
  Arms: Condition 1; Condition 11; Condition 13; Condition 15; Condition 17; Condition 19; Condition 21; Condition 23; Condition 25; Condition 27; Condition 29; Condition 3; Condition 31; Condition 5; Condition 7; Condition 9
Behavioral: Message Choice (Yes) — Participant choice drives adaptation of 1) message type delivered and 2) lapse support provision.
  Arms: Condition 10; Condition 12; Condition 14; Condition 16; Condition 18; Condition 2; Condition 20; Condition 22; Condition 24; Condition 26; Condition 28; Condition 30; Condition 32; Condition 4; Condition 6; Condition 8

SUMMARY:
Mobile obesity interventions have the potential to reach a diverse population in need; however, while effective, have not resulted in weight losses obtained in in-person interventions. Newer digital approaches called Just-in-Time Adaptive Interventions (JITAI) that offer adaptive, personalized feedback 'when needed' and in 'real time' offer an opportunity to use digital health tools "just in time". This study seeks to identify the optimal components of a comprehensive weight loss JITAI that results in weight losses that meet or exceed those in existing remotely delivered interventions.

DETAILED DESCRIPTION:
Obesity has reached epidemic proportions in the United States and is recognized as a major cause of morbidity and mortality. Young adults (18-35 years) are at particularly high risk for weight gain and obesity. In-person behavioral interventions generally produce clinically significant weight losses; however, cost and access limit their potential to reduce obesity at a population level. Although web-based interventions that mimic the structure of weekly face-to-face treatment have proven a viable alternative treatment, weight losses are generally smaller than in-person treatment. Exclusively mobile treatments have been less effective, producing 1-3 kgs over 6 months. Newer digital intervention approaches called "Just-in-Time Adaptive Interventions" (JITAIs) promise to improve upon outcomes by offering adaptive, personalized feedback on behavior "when needed" in "real time," rather than on a fixed schedule. This "just-in-time," or JIT, approach is made possible by the emergence of low-cost and widely available digital health tools that allow for the collection of continually updated health data. However, few studies have used JIT approaches in remotely delivered, fully scalable weight loss interventions. Although JITAIs are a potentially transformative approach to delivering obesity interventions, a major obstacle in their development is efficient selection of components and systematic design of an optimized intervention package that produces clinically meaningful weight losses with a population-level strategy. To solve this problem, this trial will use the Multiphase Optimization Strategy (MOST), an engineering-inspired framework, and a highly efficient experimental design to identify which levels of 5 intervention components contribute meaningfully to change in weight over 6 months among young adults with overweight and obesity. All participants (n=608) will receive a core 6-month weight loss intervention that includes evidence-based lessons, behavioral skills training, and daily weighing. With the goal of determining if greater adaptation will lead to greater weight loss, participants will be randomized to standard versus more adaptive options of 5 additional intervention components: 1) diet monitoring approach (standard vs. simplified), 2) adaptive physical activity goals (weekly vs. daily), 3) decision points for message timing (fixed vs. adaptive), 4) decision rules for message content (standard vs. adaptive), and 5) message choice (no vs. yes). Candidate components have been carefully selected from empirical evidence, tested in prior studies conducted by the research team, or in a pilot micro-randomized trial conducted by the research team. Assessments will occur at 0, 3 and 6 months to accomplish the following specific aims: 1) Build an optimized JITAI consisting of the set of intervention components that yield the greatest improvement in weight change among young adults at 6 months; 2) Conduct mediation analyses to test the relationships between the intervention components and hypothesized proximal mediators (self-regulation, competence, relatedness, relevance, autonomy) and more distal behavioral mediators (dietary intake, physical activity, and daily self-weighting); and 3) Conduct exploratory analyses of program engagement.

ELIGIBILITY:
Inclusion Criteria:

* body mass index (BMI) of 25-45 kg/m^2
* English-speaking and writing
* own a smartphone with a data and text messaging plan
* willing to be randomized to any levels of the factors

Exclusion Criteria:

* Type 1 diabetes or currently receiving medical treatment for Type 2 diabetes
* Other health problems which may influence the ability to walk for physical activity or be associated with unintentional weight change, including cancer treatment within the past 5 years or tuberculosis
* Report a heart condition, chest pain during periods of activity or rest, or loss of consciousness on the Physical Activity Readiness Questionnaire (PAR-Q; items 1-4)
* Lost 10 or more pounds (and kept it off) in the last 6 months
* Currently taking weight loss medications
* Report a past diagnosis of or current treatment for a DSM-V (Diagnostic and Statistical Manual 5) eating disorder (anorexia nervosa or bulimia nervosa)
* Currently pregnant, pregnant within the past 6 months, or planning to become pregnant within the next 6 months
* Hospitalization for depression or other psychiatric disorder within the past 12 months
* History of psychotic disorder or bipolar disorder
* Another member of the household is a participant or staff member on this trial
* Currently participating in a weight loss, nutrition or physical activity study or program or other study that would interfere with this study

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 759 (Actual)
Dates: Start 2022-04-28 (Actual); Primary Completion 2024-06-20 (Actual); Study Completion 2024-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deborah F. Tate, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred from Apr 2022 to Dec 2023; remote recruitment across the continental United States. 2510 individuals completed the online screening survey; 841 were initially eligible; out of those, 135 completed informed consent but were ineligible due to no longer being interested in participating or incomplete baseline measurement procedures, and 624 completed informed consent and all baseline assessment procedures and were randomized and enrolled in the study.
Pre-assignment Details: Individuals who signed informed consent and then completed all baseline measurement procedures (online surveys and remote weight measurements) and remained eligible were considered enrolled and were randomized to 1 of 32 conditions.
Groups:
- 1: Standard Diet Monitoring, Daily Adaptive Activity Goal, Fixed Timing, Standard Rules, No Choice: Behavioral weight loss core includes behavioral lessons, activity tracker, daily self-weighing, weekly tailored feedback summary.
  Behavioral: Standard Diet Monitoring Standard monitoring using smartphone tracking of all calorie intake.
  Behavioral: Adaptive Activity Goals (Daily) Physical activity goals that adapt once each day using the participants' data derived from activity tracker.
  Behavioral: Message Decision Points (Fixed) Message timing is fixed and evaluated at specific times each day to determine message eligibility.
  Behavioral: Message Decision Rules (Standard) Decision rules to determine eligibility to receive just-in-time messages consider participant's recent behaviors.
  Behavioral: Message Choice (No) Participant choice does not drive adaptation of 1) message type delivered or 2) lapse support provision
- 2: Standard Diet Monitoring, Daily Adaptive Activity Goal, Fixed Timing, Standard Rules, Choice: Behavioral weight loss core includes behavioral lessons, activity tracker, daily self-weighing, weekly tailored feedback summary.
  Behavioral: Standard Diet Monitoring Standard monitoring using smartphone tracking of all calorie intake.
  Behavioral: Adaptive Activity Goals (Daily) Physical activity goals that adapt once each day using the participants' data derived from activity tracker.
  Behavioral: Message Decision Points (Fixed) Message timing is fixed and evaluated at specific times each day to determine message eligibility.
  Behavioral: Message Decision Rules (Standard) Decision rules to determine eligibility to receive just-in-time messages consider participant's recent behaviors.
  Behavioral: Message Choice (Yes) Participant choice drives adaptation of 1) message type delivered and 2) lapse support provision.
- 3: Standard Diet Monitoring, Daily Adaptive Activity Goal, Fixed Timing, Adaptive Rules, No Choice: Behavioral weight loss core includes behavioral lessons, activity tracker, daily self-weighing, weekly tailored feedback summary.
  Behavioral: Standard Diet Monitoring Standard monitoring using smartphone tracking of all calorie intake.
  Behavioral: Adaptive Activity Goals (Daily) Physical activity goals that adapt once each day using the participants' data derived from activity tracker.
  Behavioral: Message Decision Points (Fixed) Message timing is fixed and evaluated at specific times each day to determine message eligibility.
  Behavioral: Message Decision Rules (Adaptive) Decision rules to determine eligibility to receive just-in-time messages consider participant's recent behaviors and overall progress.
  Behavioral: Message Choice (No) Participant choice does not drive adaptation of 1) message type delivered or 2) lapse support provision
- 4: Standard Diet Monitoring, Daily Adaptive Activity Goal, Fixed Timing, Adaptive Rules, Choice: Behavioral weight loss core includes behavioral lessons, activity tracker, daily self-weighing, weekly tailored feedback summary.
  Behavioral: Standard Diet Monitoring Standard monitoring using smartphone tracking of all calorie intake.
  Behavioral: Adaptive Activity Goals (Daily) Physical activity goals that adapt once each day using the participants' data derived from activity tracker.
  Behavioral: Message Decision Points (Fixed) Message timing is fixed and evaluated at specific times each day to determine message eligibility.
  Behavioral: Message Decision Rules (Adaptive) Decision rules to determine eligibility to receive just-in-time messages consider participant's recent behaviors and overall progress.
  Behavioral: Message Choice (Yes) Participant choice drives adaptation of 1) message type delivered and 2) lapse support provision.
- 5: Standard Diet Monitoring,Daily Adaptive Activity Goal, Adaptive Timing,Standard Rules,No Choice: Behavioral weight loss core includes behavioral lessons, activity tracker, daily self-weighing, weekly tailored feedback summary.
  Behavioral: Standard Diet Monitoring Standard monitoring using smartphone tracking of all calorie intake.
  Behavioral: Adaptive Activity Goals (Daily) Physical activity goals that adapt once each day using the participants' data derived from activity tracker.
  Behavioral: Message Decision Points (Adaptive) Message timing is adaptive and derived from individual user data to determine message eligibility.
  Behavioral: Message Decision Rules (Standard) Decision rules to determine eligibility to receive just-in-time messages consider participant's recent behaviors.
  Behavioral: Message Choice (No) Participant choice does not drive adaptation of 1) message type delivered or 2) lapse support provision
- 6: Standard Diet Monitoring, Daily Adaptive Activity Goal, Adaptive Timing, Standard Rules, Choice: Behavioral weight loss core includes behavioral lessons, activity tracker, daily self-weighing, weekly tailored feedback summary.
  Behavioral: Standard Diet Monitoring Standard monitoring using smartphone tracking of all calorie intake.
  Behavioral: Adaptive Activity Goals (Daily) Physical activity goals that adapt once each day using the participants' data derived from activity tracker.
  Behavioral: Message Decision Points (Adaptive) Message timing is adaptive and derived from individual user data to determine message eligibility.
  Behavioral: Message Decision Rules (Standard) Decision rules to determine eligibility to receive just-in-time messages consider participant's recent behaviors.
  Behavioral: Message Choice (Yes) Participant choice drives adaptation of 1) message type delivered and 2) lapse support provision.
- 7:Standard Diet Monitoring, Daily Adaptive Activity Goal, Adaptive Timing, Adaptive Rules, No Choice: Behavioral weight loss core includes behavioral lessons, activity tracker, daily self-weighing, weekly tailored feedback summary.
  Behavioral: Standard Diet Monitoring Standard monitoring using smartphone tracking of all calorie intake.
  Behavioral: Adaptive Activity Goals (Daily) Physical activity goals that adapt once each day using the participants' data derived from activity tracker.
  Behavioral: Message Decision Points (Adaptive) Message timing is adaptive and derived from individual user data to determine message eligibility.
  Behavioral: Message Decision Rules (Adaptive) Decision rules to determine eligibility to receive just-in-time messages consider participant's recent behaviors and overall progress.
  Behavioral: Message Choice (No) Participant choice does not drive adaptation of 1) message type delivered or 2) lapse support provision
- 8: Standard Diet Monitoring, Daily Adaptive Activity Goal, Adaptive Timing, Adaptive Rules, Choice: Behavioral weight loss core includes behavioral lessons, activity tracker, daily self-weighing, weekly tailored feedback summary.
  Behavioral: Standard Diet Monitoring Standard monitoring using smartphone tracking of all calorie intake.
  Behavioral: Adaptive Activity Goals (Daily) Physical activity goals that adapt once each day using the participants' data derived from activity tracker.
  Behavioral: Message Decision Points (Adaptive) Message timing is adaptive and derived from individual user data to determine message eligibility.
  Behavioral: Message Decision Rules (Adaptive) Decision rules to determine eligibility to receive just-in-time messages consider participant's recent behaviors and overall progress.
  Behavioral: Message Choice (Yes) Participant choice drives adaptation of 1) message type delivered and 2) lapse support provision.
- 9: Standard Diet Monitoring, Weekly Activity Goal, Fixed Timing, Standard Rules, No Choice: Behavioral weight loss core includes behavioral lessons, activity tracker, daily self-weighing, weekly tailored feedback summary.
  Behavioral: Standard Diet Monitoring Standard monitoring using smartphone tracking of all calorie intake.
  Behavioral: Adaptive Activity Goals (Weekly) Physical activity goals that adapt once each week using the participants' data derived from activity tracker.
  Behavioral: Message Decision Points (Fixed) Message timing is fixed and evaluated at specific times each day to determine message eligibility.
  Behavioral: Message Decision Rules (Standard) Decision rules to determine eligibility to receive just-in-time messages consider participant's recent behaviors.
  Behavioral: Message Choice (No) Participant choice does not drive adaptation of 1) message type delivered or 2) lapse support provision
- 10: Standard Diet Monitoring, Weekly Activity Goal, Fixed Timing, Standard Rules, Choice: Behavioral weight loss core includes behavioral lessons, activity tracker, daily self-weighing, weekly tailored feedback summary.
  Behavioral: Standard Diet Monitoring Standard monitoring using smartphone tracking of all calorie intake.
  Behavioral: Adaptive Activity Goals (Weekly) Physical activity goals that adapt once each week using the participants' data derived from activity tracker.
  Behavioral: Message Decision Points (Fixed) Message timing is fixed and evaluated at specific times each day to determine message eligibility.
  Behavioral: Message Decision Rules (Standard) Decision rules to determine eligibility to receive just-in-time messages consider participant's recent behaviors.
  Behavioral: Message Choice (Yes) Participant choice drives adaptation of 1) message type delivered and 2) lapse support provision.
- 11: Standard Diet Monitoring, Weekly Activity Goal, Fixed Timing, Adaptive Rules, No Choice: Behavioral weight loss core includes behavioral lessons, activity tracker, daily self-weighing, weekly tailored feedback summary.
  Behavioral: Standard Diet Monitoring Standard monitoring using smartphone tracking of all calorie intake.
  Behavioral: Adaptive Activity Goals (Weekly) Physical activity goals that adapt once each week using the participants' data derived from activity tracker.
  Behavioral: Message Decision Points (Fixed) Message timing is fixed and evaluated at specific times each day to determine message eligibility.
  Behavioral: Message Decision Rules (Adaptive) Decision rules to determine eligibility to receive just-in-time messages consider participant's recent behaviors and overall progress.
  Behavioral: Message Choice (No) Participant choice does not drive adaptation of 1) message type delivered or 2) lapse support provision
- 12: Standard Diet Monitoring, Weekly Activity Goal, Fixed Timing, Adaptive Rules, Choice: Behavioral weight loss core includes behavioral lessons, activity tracker, daily self-weighing, weekly tailored feedback summary.
  Behavioral: Standard Diet Monitoring Standard monitoring using smartphone tracking of all calorie intake.
  Behavioral: Adaptive Activity Goals (Weekly) Physical activity goals that adapt once each week using the participants' data derived from activity tracker.
  Behavioral: Message Decision Points (Fixed) Message timing is fixed and evaluated at specific times each day to determine message eligibility.
  Behavioral: Message Decision Rules (Adaptive) Decision rules to determine eligibility to receive just-in-time messages consider participant's recent behaviors and overall progress.
  Behavioral: Message Choice (Yes) Participant choice drives adaptation of 1) message type delivered and 2) lapse support provision.
- 13:Standard Diet Monitoring,Weekly Adaptive Activity Goal, Adaptive Timing, Standard Rules,No Choice: Behavioral weight loss core includes behavioral lessons, activity tracker, daily self-weighing, weekly tailored feedback summary.
  Behavioral: Standard Diet Monitoring Standard monitoring using smartphone tracking of all calorie intake.
  Behavioral: Adaptive Activity Goals (Weekly) Physical activity goals that adapt once each week using the participants' data derived from activity tracker.
  Behavioral: Message Decision Points (Adaptive) Message timing is adaptive and derived from individual user data to determine message eligibility.
  Behavioral: Message Decision Rules (Standard) Decision rules to determine eligibility to receive just-in-time messages consider participant's recent behaviors.
  Behavioral: Message Choice (No) Participant choice does not drive adaptation of 1) message type delivered or 2) lapse support provision
- 14:Standard Diet Monitoring, Weekly Adaptive Activity Goal, Adaptive Timing, Standard Rules, Choice: Behavioral weight loss core includes behavioral lessons, activity tracker, daily self-weighing, weekly tailored feedback summary.
  Behavioral: Standard Diet Monitoring Standard monitoring using smartphone tracking of all calorie intake.
  Behavioral: Adaptive Activity Goals (Weekly) Physical activity goals that adapt once each week using the participants' data derived from activity tracker.
  Behavioral: Message Decision Points (Adaptive) Message timing is adaptive and derived from individual user data to determine message eligibility.
  Behavioral: Message Decision Rules (Standard) Decision rules to determine eligibility to receive just-in-time messages consider participant's recent behaviors.
  Behavioral: Message Choice (Yes) Participant choice drives adaptation of 1) message type delivered and 2) lapse support provision.
- 15:Standard Diet Monitoring,Weekly Adaptive Activity Goal,Adaptive Timing, Adaptive Rules, No Choice: Behavioral weight loss core includes behavioral lessons, activity tracker, daily self-weighing, weekly tailored feedback summary.
  Behavioral: Standard Diet Monitoring Standard monitoring using smartphone tracking of all calorie intake.
  Behavioral: Adaptive Activity Goals (Weekly) Physical activity goals that adapt once each week using the participants' data derived from activity tracker.
  Behavioral: Message Decision Points (Adaptive) Message timing is adaptive and derived from individual user data to determine message eligibility.
  Behavioral: Message Decision Rules (Adaptive) Decision rules to determine eligibility to receive just-in-time messages consider participant's recent behaviors and overall progress.
  Behavioral: Message Choice (No) Participant choice does not drive adaptation of 1) message type delivered or 2) lapse support provision
- 16: Standard Diet Monitoring, Weekly Adaptive Activity Goal, Adaptive Timing, Adaptive Rules, Choice: Behavioral weight loss core includes behavioral lessons, activity tracker, daily self-weighing, weekly tailored feedback summary.
  Behavioral: Standard Diet Monitoring Standard monitoring using smartphone tracking of all calorie intake.
  Behavioral: Adaptive Activity Goals (Weekly) Physical activity goals that adapt once each week using the participants' data derived from activity tracker.
  Behavioral: Message Decision Points (Adaptive) Message timing is adaptive and derived from individual user data to determine message eligibility.
  Behavioral: Message Decision Rules (Adaptive) Decision rules to determine eligibility to receive just-in-time messages consider participant's recent behaviors and overall progress.
  Behavioral: Message Choice (Yes) Participant choice drives adaptation of 1) message type delivered and 2) lapse support provision.
- 17:Simplified Diet Monitoring, Daily Adaptive Activity Goal, Fixed Timing, Standard Rules, No Choice: Behavioral weight loss core includes behavioral lessons, activity tracker, daily self-weighing, weekly tailored feedback summary.
  Behavioral: Simplified Diet Monitoring Simplified diet monitoring using smartphone tracking of red foods using a traffic light approach.
  Behavioral: Adaptive Activity Goals (Daily) Physical activity goals that adapt once each day using the participants' data derived from activity tracker.
  Behavioral: Message Decision Points (Fixed) Message timing is fixed and evaluated at specific times each day to determine message eligibility.
  Behavioral: Message Decision Rules (Standard) Decision rules to determine eligibility to receive just-in-time messages consider participant's recent behaviors.
  Behavioral: Message Choice (No) Participant choice does not drive adaptation of 1) message type delivered or 2) lapse support provision
- 18: Simplified Diet Monitoring, Daily Adaptive Activity Goal, Fixed Timing, Standard Rules, Choice: Behavioral weight loss core includes behavioral lessons, activity tracker, daily self-weighing, weekly tailored feedback summary.
  Behavioral: Simplified Diet Monitoring Simplified diet monitoring using smartphone tracking of red foods using a traffic light approach.
  Behavioral: Adaptive Activity Goals (Daily) Physical activity goals that adapt once each day using the participants' data derived from activity tracker.
  Behavioral: Message Decision Points (Fixed) Message timing is fixed and evaluated at specific times each day to determine message eligibility.
  Behavioral: Message Decision Rules (Standard) Decision rules to determine eligibility to receive just-in-time messages consider participant's recent behaviors.
  Behavioral: Message Choice (Yes) Participant choice drives adaptation of 1) message type delivered and 2) lapse support provision.
- 19:Simplified Diet Monitoring, Daily Adaptive Activity Goal, Fixed Timing, Adaptive Rules, No Choice: Behavioral weight loss core includes behavioral lessons, activity tracker, daily self-weighing, weekly tailored feedback summary.
  Behavioral: Simplified Diet Monitoring Simplified diet monitoring using smartphone tracking of red foods using a traffic light approach.
  Behavioral: Adaptive Activity Goals (Daily) Physical activity goals that adapt once each day using the participants' data derived from activity tracker.
  Behavioral: Message Decision Points (Fixed) Message timing is fixed and evaluated at specific times each day to determine message eligibility.
  Behavioral: Message Decision Rules (Adaptive) Decision rules to determine eligibility to receive just-in-time messages consider participant's recent behaviors and overall progress.
  Behavioral: Message Choice (No) Participant choice does not drive adaptation of 1) message type delivered or 2) lapse support provision
- 20: Simplified Diet Monitoring, Daily Adaptive Activity Goal, Fixed Timing, Adaptive Rules, Choice: Behavioral weight loss core includes behavioral lessons, activity tracker, daily self-weighing, weekly tailored feedback summary.
  Behavioral: Simplified Diet Monitoring Simplified diet monitoring using smartphone tracking of red foods using a traffic light approach.
  Behavioral: Adaptive Activity Goals (Daily) Physical activity goals that adapt once each day using the participants' data derived from activity tracker.
  Behavioral: Message Decision Points (Fixed) Message timing is fixed and evaluated at specific times each day to determine message eligibility.
  Behavioral: Message Decision Rules (Adaptive) Decision rules to determine eligibility to receive just-in-time messages consider participant's recent behaviors and overall progress.
  Behavioral: Message Choice (Yes) Participant choice drives adaptation of 1) message type delivered and 2) lapse support provision.
- 21:Simplified Diet Monitoring,Daily Adaptive Activity Goal,Adaptive Timing,Standard Rules, No Choice: Behavioral weight loss core includes behavioral lessons, activity tracker, daily self-weighing, weekly tailored feedback summary.
  Behavioral: Simplified Diet Monitoring Simplified diet monitoring using smartphone tracking of red foods using a traffic light approach.
  Behavioral: Adaptive Activity Goals (Daily) Physical activity goals that adapt once each day using the participants' data derived from activity tracker.
  Behavioral: Message Decision Points (Adaptive) Message timing is adaptive and derived from individual user data to determine message eligibility.
  Behavioral: Message Decision Rules (Standard) Decision rules to determine eligibility to receive just-in-time messages consider participant's recent behaviors.
  Behavioral: Message Choice (No) Participant choice does not drive adaptation of 1) message type delivered or 2) lapse support provision
- 22:Simplified Diet Monitoring, Daily Adaptive Activity Goal, Adaptive Timing, Standard Rules, Choice: Behavioral weight loss core includes behavioral lessons, activity tracker, daily self-weighing, weekly tailored feedback summary.
  Behavioral: Simplified Diet Monitoring Simplified diet monitoring using smartphone tracking of red foods using a traffic light approach.
  Behavioral: Adaptive Activity Goals (Daily) Physical activity goals that adapt once each day using the participants' data derived from activity tracker.
  Behavioral: Message Decision Points (Adaptive) Message timing is adaptive and derived from individual user data to determine message eligibility.
  Behavioral: Message Decision Rules (Standard) Decision rules to determine eligibility to receive just-in-time messages consider participant's recent behaviors.
  Behavioral: Message Choice (Yes) Participant choice drives adaptation of 1) message type delivered and 2) lapse support provision.
- 23:Simplified Diet Monitoring,Daily Adaptive Activity Goal,Adaptive Timing,Adaptive Rules, No Choice: Behavioral weight loss core includes behavioral lessons, activity tracker, daily self-weighing, weekly tailored feedback summary.
  Behavioral: Simplified Diet Monitoring Simplified diet monitoring using smartphone tracking of red foods using a traffic light approach.
  Behavioral: Adaptive Activity Goals (Daily) Physical activity goals that adapt once each day using the participants' data derived from activity tracker.
  Behavioral: Message Decision Points (Adaptive) Message timing is adaptive and derived from individual user data to determine message eligibility.
  Behavioral: Message Decision Rules (Adaptive) Decision rules to determine eligibility to receive just-in-time messages consider participant's recent behaviors and overall progress.
  Behavioral: Message Choice (No) Participant choice does not drive adaptation of 1) message type delivered or 2) lapse support provision
- 24:Simplified Diet Monitoring, Daily Adaptive Activity Goal, Adaptive Timing, Adaptive Rules, Choice: Behavioral weight loss core includes behavioral lessons, activity tracker, daily self-weighing, weekly tailored feedback summary.
  Behavioral: Simplified Diet Monitoring Simplified diet monitoring using smartphone tracking of red foods using a traffic light approach.
  Behavioral: Adaptive Activity Goals (Daily) Physical activity goals that adapt once each day using the participants' data derived from activity tracker.
  Behavioral: Message Decision Points (Adaptive) Message timing is adaptive and derived from individual user data to determine message eligibility.
  Behavioral: Message Decision Rules (Adaptive) Decision rules to determine eligibility to receive just-in-time messages consider participant's recent behaviors and overall progress.
  Behavioral: Message Choice (Yes) Participant choice drives adaptation of 1) message type delivered and 2) lapse support provision.
- 25:Simplified Diet Monitoring,Weekly Adaptive Activity Goal, Fixed Timing, Standard Rules, No Choice: Behavioral weight loss core includes behavioral lessons, activity tracker, daily self-weighing, weekly tailored feedback summary.
  Behavioral: Simplified Diet Monitoring Simplified diet monitoring using smartphone tracking of red foods using a traffic light approach.
  Behavioral: Adaptive Activity Goals (Weekly) Physical activity goals that adapt once each week using the participants' data derived from activity tracker.
  Behavioral: Message Decision Points (Fixed) Message timing is fixed and evaluated at specific times each day to determine message eligibility.
  Behavioral: Message Decision Rules (Standard) Decision rules to determine eligibility to receive just-in-time messages consider participant's recent behaviors.
  Behavioral: Message Choice (No) Participant choice does not drive adaptation of 1) message type delivered or 2) lapse support provision
- 26: Simplified Diet Monitoring, Weekly Adaptive Activity Goal, Fixed Timing, Standard Rules, Choice: Behavioral weight loss core includes behavioral lessons, activity tracker, daily self-weighing, weekly tailored feedback summary.
  Behavioral: Simplified Diet Monitoring Simplified diet monitoring using smartphone tracking of red foods using a traffic light approach.
  Behavioral: Adaptive Activity Goals (Weekly) Physical activity goals that adapt once each week using the participants' data derived from activity tracker.
  Behavioral: Message Decision Points (Fixed) Message timing is fixed and evaluated at specific times each day to determine message eligibility.
  Behavioral: Message Decision Rules (Standard) Decision rules to determine eligibility to receive just-in-time messages consider participant's recent behaviors.
  Behavioral: Message Choice (Yes) Participant choice drives adaptation of 1) message type delivered and 2) lapse support provision.
- 27:Simplified Diet Monitoring,Weekly Adaptive Activity Goal, Fixed Timing, Adaptive Rules, No Choice: Behavioral weight loss core includes behavioral lessons, activity tracker, daily self-weighing, weekly tailored feedback summary.
  Behavioral: Simplified Diet Monitoring Simplified diet monitoring using smartphone tracking of red foods using a traffic light approach.
  Behavioral: Adaptive Activity Goals (Weekly) Physical activity goals that adapt once each week using the participants' data derived from activity tracker.
  Behavioral: Message Decision Points (Fixed) Message timing is fixed and evaluated at specific times each day to determine message eligibility.
  Behavioral: Message Decision Rules (Adaptive) Decision rules to determine eligibility to receive just-in-time messages consider participant's recent behaviors and overall progress.
  Behavioral: Message Choice (No) Participant choice does not drive adaptation of 1) message type delivered or 2) lapse support provision
- 28: Simplified Diet Monitoring, Weekly Adaptive Activity Goal, Fixed Timing, Adaptive Rules, Choice: Behavioral weight loss core includes behavioral lessons, activity tracker, daily self-weighing, weekly tailored feedback summary.
  Behavioral: Simplified Diet Monitoring Simplified diet monitoring using smartphone tracking of red foods using a traffic light approach.
  Behavioral: Adaptive Activity Goals (Weekly) Physical activity goals that adapt once each week using the participants' data derived from activity tracker.
  Behavioral: Message Decision Points (Fixed) Message timing is fixed and evaluated at specific times each day to determine message eligibility.
  Behavioral: Message Decision Rules (Adaptive) Decision rules to determine eligibility to receive just-in-time messages consider participant's recent behaviors and overall progress.
  Behavioral: Message Choice (Yes) Participant choice drives adaptation of 1) message type delivered and 2) lapse support provision.
- 29:Simplified Diet Monitoring,Weekly Adaptive Activity Goal,Adaptive Timing,Standard Rules,No Choice: Behavioral weight loss core includes behavioral lessons, activity tracker, daily self-weighing, weekly tailored feedback summary.
  Behavioral: Simplified Diet Monitoring Simplified diet monitoring using smartphone tracking of red foods using a traffic light approach.
  Behavioral: Adaptive Activity Goals (Weekly) Physical activity goals that adapt once each week using the participants' data derived from activity tracker.
  Behavioral: Message Decision Points (Adaptive) Message timing is adaptive and derived from individual user data to determine message eligibility.
  Behavioral: Message Decision Rules (Standard) Decision rules to determine eligibility to receive just-in-time messages consider participant's recent behaviors.
  Behavioral: Message Choice (No) Participant choice does not drive adaptation of 1) message type delivered or 2) lapse support provision
- 30:Simplified Diet Monitoring,Weekly Adaptive Activity Goal, Adaptive Timing, Standard Rules, Choice: Behavioral weight loss core includes behavioral lessons, activity tracker, daily self-weighing, weekly tailored feedback summary.
  Behavioral: Simplified Diet Monitoring Simplified diet monitoring using smartphone tracking of red foods using a traffic light approach.
  Behavioral: Adaptive Activity Goals (Weekly) Physical activity goals that adapt once each week using the participants' data derived from activity tracker.
  Behavioral: Message Decision Points (Adaptive) Message timing is adaptive and derived from individual user data to determine message eligibility.
  Behavioral: Message Decision Rules (Standard) Decision rules to determine eligibility to receive just-in-time messages consider participant's recent behaviors.
  Behavioral: Message Choice (Yes) Participant choice drives adaptation of 1) message type delivered and 2) lapse support provision.
- 31:Simplified Diet Monitoring,Weekly Adaptive Activity Goal,Adaptive Timing,Adaptive Rules,No Choice: Behavioral weight loss core includes behavioral lessons, activity tracker, daily self-weighing, weekly tailored feedback summary.
  Behavioral: Simplified Diet Monitoring Simplified diet monitoring using smartphone tracking of red foods using a traffic light approach.
  Behavioral: Adaptive Activity Goals (Weekly) Physical activity goals that adapt once each week using the participants' data derived from activity tracker.
  Behavioral: Message Decision Points (Adaptive) Message timing is adaptive and derived from individual user data to determine message eligibility.
  Behavioral: Message Decision Rules (Adaptive) Decision rules to determine eligibility to receive just-in-time messages consider participant's recent behaviors and overall progress.
  Behavioral: Message Choice (No) Participant choice does not drive adaptation of 1) message type delivered or 2) lapse support provision
- 32:Simplified Diet Monitoring, Weekly Adaptive Activity Goal, Adaptive Timing, Adaptive Rules,Choice: Behavioral weight loss core includes behavioral lessons, activity tracker, daily self-weighing, weekly tailored feedback summary.
  Behavioral: Simplified Diet Monitoring Simplified diet monitoring using smartphone tracking of red foods using a traffic light approach.
  Behavioral: Adaptive Activity Goals (Weekly) Physical activity goals that adapt once each week using the participants' data derived from activity tracker.
  Behavioral: Message Decision Points (Adaptive) Message timing is adaptive and derived from individual user data to determine message eligibility.
  Behavioral: Message Decision Rules (Adaptive) Decision rules to determine eligibility to receive just-in-time messages consider participant's recent behaviors and overall progress.
  Behavioral: Message Choice (Yes) Participant choice drives adaptation of 1) message type delivered and 2) lapse support provision.
Period: Overall Study
Arm/Group | 1: Standard Diet Monitoring, Daily Adaptive Activity Goal, Fixed Timing, Standard Rules, No Choice | 2: Standard Diet Monitoring, Daily Adaptive Activity Goal, Fixed Timing, Standard Rules, Choice | 3: Standard Diet Monitoring, Daily Adaptive Activity Goal, Fixed Timing, Adaptive Rules, No Choice | 4: Standard Diet Monitoring, Daily Adaptive Activity Goal, Fixed Timing, Adaptive Rules, Choice | 5: Standard Diet Monitoring,Daily Adaptive Activity Goal, Adaptive Timing,Standard Rules,No Choice | 6: Standard Diet Monitoring, Daily Adaptive Activity Goal, Adaptive Timing, Standard Rules, Choice | 7:Standard Diet Monitoring, Daily Adaptive Activity Goal, Adaptive Timing, Adaptive Rules, No Choice | 8: Standard Diet Monitoring, Daily Adaptive Activity Goal, Adaptive Timing, Adaptive Rules, Choice | 9: Standard Diet Monitoring, Weekly Activity Goal, Fixed Timing, Standard Rules, No Choice | 10: Standard Diet Monitoring, Weekly Activity Goal, Fixed Timing, Standard Rules, Choice | 11: Standard Diet Monitoring, Weekly Activity Goal, Fixed Timing, Adaptive Rules, No Choice | 12: Standard Diet Monitoring, Weekly Activity Goal, Fixed Timing, Adaptive Rules, Choice | 13:Standard Diet Monitoring,Weekly Adaptive Activity Goal, Adaptive Timing, Standard Rules,No Choice | 14:Standard Diet Monitoring, Weekly Adaptive Activity Goal, Adaptive Timing, Standard Rules, Choice | 15:Standard Diet Monitoring,Weekly Adaptive Activity Goal,Adaptive Timing, Adaptive Rules, No Choice | 16: Standard Diet Monitoring, Weekly Adaptive Activity Goal, Adaptive Timing, Adaptive Rules, Choice | 17:Simplified Diet Monitoring, Daily Adaptive Activity Goal, Fixed Timing, Standard Rules, No Choice | 18: Simplified Diet Monitoring, Daily Adaptive Activity Goal, Fixed Timing, Standard Rules, Choice | 19:Simplified Diet Monitoring, Daily Adaptive Activity Goal, Fixed Timing, Adaptive Rules, No Choice | 20: Simplified Diet Monitoring, Daily Adaptive Activity Goal, Fixed Timing, Adaptive Rules, Choice | 21:Simplified Diet Monitoring,Daily Adaptive Activity Goal,Adaptive Timing,Standard Rules, No Choice | 22:Simplified Diet Monitoring, Daily Adaptive Activity Goal, Adaptive Timing, Standard Rules, Choice | 23:Simplified Diet Monitoring,Daily Adaptive Activity Goal,Adaptive Timing,Adaptive Rules, No Choice | 24:Simplified Diet Monitoring, Daily Adaptive Activity Goal, Adaptive Timing, Adaptive Rules, Choice | 25:Simplified Diet Monitoring,Weekly Adaptive Activity Goal, Fixed Timing, Standard Rules, No Choice | 26: Simplified Diet Monitoring, Weekly Adaptive Activity Goal, Fixed Timing, Standard Rules, Choice | 27:Simplified Diet Monitoring,Weekly Adaptive Activity Goal, Fixed Timing, Adaptive Rules, No Choice | 28: Simplified Diet Monitoring, Weekly Adaptive Activity Goal, Fixed Timing, Adaptive Rules, Choice | 29:Simplified Diet Monitoring,Weekly Adaptive Activity Goal,Adaptive Timing,Standard Rules,No Choice | 30:Simplified Diet Monitoring,Weekly Adaptive Activity Goal, Adaptive Timing, Standard Rules, Choice | 31:Simplified Diet Monitoring,Weekly Adaptive Activity Goal,Adaptive Timing,Adaptive Rules,No Choice | 32:Simplified Diet Monitoring, Weekly Adaptive Activity Goal, Adaptive Timing, Adaptive Rules,Choice
Started | 18 | 21 | 20 | 18 | 20 | 18 | 19 | 20 | 20 | 20 | 20 | 19 | 18 | 19 | 20 | 19 | 20 | 20 | 20 | 19 | 20 | 19 | 20 | 19 | 19 | 20 | 20 | 20 | 20 | 20 | 20 | 19
Completed 3-Month Visit | 17 | 20 | 20 | 18 | 20 | 18 | 19 | 20 | 20 | 20 | 20 | 19 | 18 | 19 | 20 | 19 | 20 | 19 | 19 | 19 | 19 | 19 | 20 | 19 | 19 | 20 | 19 | 20 | 20 | 20 | 19 | 19
Completed | 17 | 20 | 18 | 18 | 20 | 16 | 19 | 17 | 19 | 18 | 18 | 18 | 16 | 18 | 18 | 19 | 20 | 17 | 18 | 18 | 18 | 19 | 18 | 16 | 19 | 18 | 19 | 20 | 19 | 20 | 17 | 18
Not Completed | 1 | 1 | 2 | 0 | 0 | 2 | 0 | 3 | 1 | 2 | 2 | 1 | 2 | 1 | 2 | 0 | 0 | 3 | 2 | 1 | 2 | 0 | 2 | 3 | 0 | 2 | 1 | 0 | 1 | 0 | 3 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 1 | 0 | 2 | 0 | 0 | 2 | 0 | 1 | 1 | 2 | 2 | 1 | 1 | 0 | 1 | 0 | 0 | 2 | 1 | 0 | 1 | 0 | 2 | 1 | 0 | 2 | 0 | 0 | 1 | 0 | 2 | 1

BASELINE CHARACTERISTICS:
Population: Baseline population included all randomized participants, N=624.
Groups:
- Total: Total of all reporting groups
Arm/Group | 1: Standard Diet Monitoring, Daily Adaptive Activity Goal, Fixed Timing, Standard Rules, No Choice | 2: Standard Diet Monitoring, Daily Adaptive Activity Goal, Fixed Timing, Standard Rules, Choice | 3: Standard Diet Monitoring, Daily Adaptive Activity Goal, Fixed Timing, Adaptive Rules, No Choice | 4: Standard Diet Monitoring, Daily Adaptive Activity Goal, Fixed Timing, Adaptive Rules, Choice | 5: Standard Diet Monitoring,Daily Adaptive Activity Goal, Adaptive Timing,Standard Rules,No Choice | 6: Standard Diet Monitoring, Daily Adaptive Activity Goal, Adaptive Timing, Standard Rules, Choice | 7:Standard Diet Monitoring, Daily Adaptive Activity Goal, Adaptive Timing, Adaptive Rules, No Choice | 8: Standard Diet Monitoring, Daily Adaptive Activity Goal, Adaptive Timing, Adaptive Rules, Choice | 9: Standard Diet Monitoring, Weekly Activity Goal, Fixed Timing, Standard Rules, No Choice | 10: Standard Diet Monitoring, Weekly Activity Goal, Fixed Timing, Standard Rules, Choice | 11: Standard Diet Monitoring, Weekly Activity Goal, Fixed Timing, Adaptive Rules, No Choice | 12: Standard Diet Monitoring, Weekly Activity Goal, Fixed Timing, Adaptive Rules, Choice | 13:Standard Diet Monitoring,Weekly Adaptive Activity Goal, Adaptive Timing, Standard Rules,No Choice | 14:Standard Diet Monitoring, Weekly Adaptive Activity Goal, Adaptive Timing, Standard Rules, Choice | 15:Standard Diet Monitoring,Weekly Adaptive Activity Goal,Adaptive Timing, Adaptive Rules, No Choice | 16: Standard Diet Monitoring, Weekly Adaptive Activity Goal, Adaptive Timing, Adaptive Rules, Choice | 17:Simplified Diet Monitoring, Daily Adaptive Activity Goal, Fixed Timing, Standard Rules, No Choice | 18: Simplified Diet Monitoring, Daily Adaptive Activity Goal, Fixed Timing, Standard Rules, Choice | 19:Simplified Diet Monitoring, Daily Adaptive Activity Goal, Fixed Timing, Adaptive Rules, No Choice | 20: Simplified Diet Monitoring, Daily Adaptive Activity Goal, Fixed Timing, Adaptive Rules, Choice | 21:Simplified Diet Monitoring,Daily Adaptive Activity Goal,Adaptive Timing,Standard Rules, No Choice | 22:Simplified Diet Monitoring, Daily Adaptive Activity Goal, Adaptive Timing, Standard Rules, Choice | 23:Simplified Diet Monitoring,Daily Adaptive Activity Goal,Adaptive Timing,Adaptive Rules, No Choice | 24:Simplified Diet Monitoring, Daily Adaptive Activity Goal, Adaptive Timing, Adaptive Rules, Choice | 25:Simplified Diet Monitoring,Weekly Adaptive Activity Goal, Fixed Timing, Standard Rules, No Choice | 26: Simplified Diet Monitoring, Weekly Adaptive Activity Goal, Fixed Timing, Standard Rules, Choice | 27:Simplified Diet Monitoring,Weekly Adaptive Activity Goal, Fixed Timing, Adaptive Rules, No Choice | 28: Simplified Diet Monitoring, Weekly Adaptive Activity Goal, Fixed Timing, Adaptive Rules, Choice | 29:Simplified Diet Monitoring,Weekly Adaptive Activity Goal,Adaptive Timing,Standard Rules,No Choice | 30:Simplified Diet Monitoring,Weekly Adaptive Activity Goal, Adaptive Timing, Standard Rules, Choice | 31:Simplified Diet Monitoring,Weekly Adaptive Activity Goal,Adaptive Timing,Adaptive Rules,No Choice | 32:Simplified Diet Monitoring, Weekly Adaptive Activity Goal, Adaptive Timing, Adaptive Rules,Choice | Total
Number analyzed (Participants) | 18 | 21 | 20 | 18 | 20 | 18 | 19 | 20 | 20 | 20 | 20 | 19 | 18 | 19 | 20 | 19 | 20 | 20 | 20 | 19 | 20 | 19 | 20 | 19 | 19 | 20 | 20 | 20 | 20 | 20 | 20 | 19 | 624
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.4 (5.6) | 30.9 (5.4) | 33.2 (4.4) | 31.4 (5.0) | 31.3 (4.6) | 32.1 (4.5) | 29.0 (4.7) | 29.9 (5.7) | 30.1 (4.7) | 33.5 (4.0) | 30.6 (4.7) | 32.4 (4.9) | 30.3 (3.2) | 32.4 (4.5) | 32.8 (3.9) | 31.2 (5.7) | 30.9 (4.5) | 30.0 (5.3) | 29.5 (5.3) | 30.5 (4.9) | 31.4 (4.3) | 30.9 (4.8) | 30.5 (6.0) | 27.1 (5.4) | 33.0 (3.9) | 30.7 (6.2) | 32.9 (3.8) | 31.2 (4.7) | 31.2 (5.0) | 32.6 (4.5) | 29.7 (4.9) | 33.6 (4.1) | 31.2 (4.9)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 13 | 14 | 11 | 12 | 10 | 9 | 14 | 14 | 14 | 16 | 16 | 11 | 12 | 9 | 13 | 11 | 14 | 15 | 14 | 16 | 14 | 14 | 10 | 14 | 14 | 14 | 16 | 13 | 12 | 12 | 13 | 14 | 418
  Male | 4 | 7 | 9 | 6 | 9 | 8 | 5 | 6 | 6 | 4 | 4 | 8 | 6 | 10 | 7 | 8 | 6 | 5 | 6 | 3 | 6 | 5 | 10 | 5 | 5 | 6 | 4 | 7 | 8 | 8 | 7 | 5 | 203
  Don't know | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Prefer not to answer | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 3 | 3 | 2 | 1 | 1 | 3 | 6 | 3 | 1 | 3 | 4 | 1 | 3 | 1 | 1 | 3 | 3 | 1 | 0 | 5 | 3 | 2 | 2 | 2 | 4 | 1 | 5 | 4 | 1 | 2 | 79
  Not Hispanic or Latino | 15 | 18 | 16 | 15 | 17 | 17 | 18 | 17 | 14 | 16 | 19 | 16 | 14 | 18 | 17 | 18 | 19 | 17 | 17 | 16 | 20 | 13 | 17 | 17 | 17 | 18 | 16 | 19 | 15 | 16 | 18 | 17 | 537
  Unknown or Not Reported | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 4
  Asian | 4 | 1 | 2 | 0 | 2 | 5 | 2 | 1 | 2 | 1 | 4 | 2 | 2 | 4 | 0 | 5 | 4 | 4 | 1 | 2 | 2 | 1 | 6 | 1 | 0 | 3 | 1 | 3 | 2 | 3 | 3 | 0 | 73
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 7 | 2 | 3 | 4 | 2 | 2 | 4 | 3 | 4 | 6 | 1 | 2 | 5 | 3 | 5 | 4 | 6 | 3 | 5 | 4 | 4 | 3 | 3 | 6 | 2 | 7 | 2 | 4 | 1 | 5 | 8 | 122
  White | 8 | 11 | 12 | 13 | 13 | 9 | 14 | 15 | 14 | 11 | 8 | 15 | 11 | 10 | 15 | 9 | 10 | 8 | 12 | 7 | 13 | 10 | 10 | 13 | 10 | 14 | 8 | 14 | 12 | 13 | 10 | 9 | 361
  More than one race | 2 | 2 | 2 | 1 | 0 | 2 | 0 | 0 | 1 | 2 | 1 | 1 | 3 | 0 | 2 | 0 | 1 | 1 | 2 | 3 | 1 | 2 | 1 | 1 | 0 | 1 | 4 | 0 | 1 | 2 | 0 | 1 | 40
  Unknown or Not Reported | 2 | 0 | 2 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 2 | 0 | 2 | 0 | 1 | 2 | 0 | 0 | 1 | 1 | 1 | 2 | 0 | 24
Weight (lb) [Mean (Standard Deviation); unit: pounds] | 207.7 (52.3) | 208.5 (35.1) | 206.8 (45.1) | 214.9 (38.7) | 210.5 (41.5) | 212.1 (36.3) | 195.7 (36.5) | 200.3 (43.3) | 203.1 (33.4) | 208.8 (33.2) | 195.2 (32.4) | 224.4 (36.2) | 190.8 (28.5) | 233.9 (45.6) | 218.2 (39.8) | 185.7 (34.3) | 200.7 (49.7) | 195.0 (47.7) | 219.5 (53.4) | 201.5 (41.8) | 206.1 (36.3) | 211.0 (39.6) | 207.5 (45.6) | 216.3 (45.1) | 210.6 (33.6) | 203.8 (40.4) | 203.0 (37.1) | 200.9 (33.9) | 218.3 (42.0) | 198.5 (22.3) | 206.0 (49.8) | 215.8 (33.5) | 207.2 (40.3)

OUTCOME MEASURES:

1. Primary Outcome: Weight (kg)
Description: Estimated mean weight change in kg from baseline to 6 months for each of the two levels of each component (factor) obtained from intent-to-treat (ITT) linear mixed models of analysis of variance. More negative values of weight change indicate greater weight loss (6-month weight - baseline weight).
Time Frame: Baseline, 6 months
Population: ITT: all randomized participants using all available weights.
Measure: Mean (95% Confidence Interval); unit: kg
Groups:
- Weekly Adaptive Activity Goals: Physical activity goals that adapt once each week using the participants' data derived from activity tracker.
- Daily Adaptive Activity Goals: Physical activity goals that adapt once each day using the participants' data derived from activity tracker.
- Fixed Message Decision Points: Message timing is fixed and evaluated at specific times each day to determine message eligibility.
- Adaptive Message Decision Points: Message timing is adaptive and derived from individual user data to determine message eligibility.
- Standard Message Decision Rules: Decision rules to determine eligibility to receive just-in-time messages consider participant's recent behaviors.
- Adaptive Message Decision Rules: Decision rules to determine eligibility to receive just-in-time messages consider participant's recent behaviors and overall progress.
- No Message Choice: Participant choice does not drive adaptation of 1) message type delivered or 2) lapse support provision
- Message Choice: Participant choice drives adaptation of 1) message type delivered and 2) lapse support provision.
Arm/Group | Standard Diet Monitoring | Simplified Diet Monitoring | Weekly Adaptive Activity Goals | Daily Adaptive Activity Goals | Fixed Message Decision Points | Adaptive Message Decision Points | Standard Message Decision Rules | Adaptive Message Decision Rules | No Message Choice | Message Choice
Number analyzed (Participants) | 309 | 315 | 313 | 311 | 314 | 310 | 312 | 312 | 314 | 310
kg | -3.61 [-4.25 to -2.97] | -3.31 [-3.95 to -2.68] | -3.32 [-3.96 to -2.68] | -3.60 [-4.24 to -2.96] | -3.66 [-4.29 to -3.02] | -3.26 [-3.90 to -2.61] | -3.65 [-4.29 to -3.02] | -3.26 [-3.91 to -2.62] | -3.19 [-3.83 to -2.55] | -3.73 [-4.38 to -3.09]
Statistical Analysis 1: Comparison: Standard Diet Monitoring vs Simplified Diet Monitoring; ITT analysis for factor 1 (dietary self-monitoring) using linear mixed models comparing the effect of standard dietary monitoring to simplified dietary monitoring on weight change over time (from baseline to 6 months); Test type: Superiority; p = 0.52, Mixed Models Analysis; Degrees of freedom (2,622); Mean Difference (Net) = 0.30, 95% CI 2-sided [-0.61 to 1.20] — Standard dietary monitoring coded as 0 (reference) and simplified dietary monitoring coded as 1; a positive estimation parameter indicates that the reference group had greater (more negative) weight loss
Statistical Analysis 2: Comparison: Weekly Adaptive Activity Goals vs Daily Adaptive Activity Goals; ITT analysis for factor 2 (adaptive activity goals) using linear mixed models comparing the effect of weekly adaptive activity goals versus daily adaptive activity goals on weight change over time (from baseline to 6 months); Test type: Superiority; p = 0.54, Mixed Models Analysis; Degrees of freedom (2,622); Mean Difference (Net) = -0.28, 95% CI 2-sided [-1.19 to 0.63] — Weekly adaptive goals coded as 0 (reference) and daily adaptive goals coded as 1; a positive estimation parameter indicates that the reference group had greater (more negative) weight loss
Statistical Analysis 3: Comparison: Fixed Message Decision Points vs Adaptive Message Decision Points; ITT analysis for factor 3 (message decision points) using linear mixed models comparing the effect of weekly adaptive activity goals versus daily adaptive activity goals on weight change over time (from baseline to 6 months); Test type: Superiority; p = 0.39, Mixed Models Analysis; Degrees of freedom (2,622); Mean Difference (Net) = 0.40, 95% CI 2-sided [-0.50 to 1.31] — Fixed message decision points coded as 0 (reference) and adaptive message decision points coded as 1; a positive estimation parameter indicates that the reference group had greater (more negative) weight loss
Statistical Analysis 4: Comparison: Standard Message Decision Rules vs Adaptive Message Decision Rules; ITT analysis for factor 4 (message decision rules) using linear mixed models comparing the effect of standard decision rules to adaptive decision rules on weight change over time (from baseline to 6 months); Test type: Superiority; p = 0.70, Mixed Models Analysis; Degrees of freedom (2,622); Mean Difference (Net) = 0.39, 95% CI 2-sided [-0.52 to 1.30] — Standard decision rules coded as 0 (reference) and adaptive decision rules coded as 1; a positive estimation parameter indicates that the reference group had greater (more negative) weight loss
Statistical Analysis 5: Comparison: No Message Choice vs Message Choice; ITT analysis for factor 5 (participant choice) using linear mixed models comparing the effect of no participant message choice versus participant message choice on weight change over time (from baseline to 6 months); Test type: Superiority; p = 0.47, Mixed Models Analysis; Degrees of freedom (2,622); Mean Difference (Net) = -0.55, 95% CI 2-sided [-1.45 to 0.36] — No choice points coded as 0 (reference) and Choice coded as 1; a positive estimation parameter indicates that the reference group had greater (more negative) weight loss

2. Secondary Outcome: Weight (kg)
Description: Estimated mean weight change in kg from baseline to 3 months for each of the two levels of each component (factor) obtained from intent-to-treat (ITT) linear mixed models of analysis of variance. More negative values of weight change indicate greater weight loss (3-month weight - baseline weight).
Time Frame: Baseline, 3 months
Measure: Mean (95% Confidence Interval); unit: kg
Arm/Group | Standard Diet Monitoring | Simplified Diet Monitoring | Weekly Adaptive Activity Goals | Daily Adaptive Activity Goals | Fixed Message Decision Points | Adaptive Message Decision Points | Standard Message Decision Rules | Adaptive Message Decision Rules | No Message Choice | Message Choice
Number analyzed (Participants) | 309 | 315 | 313 | 311 | 314 | 310 | 312 | 312 | 314 | 310
kg | -2.54 [-2.97 to -2.12] | -2.30 [-2.72 to -1.88] | -2.22 [-2.64 to -1.80] | -2.63 [-3.06 to -2.21] | -2.69 [-3.11 to -2.27] | -2.16 [-2.58 to -1.74] | -2.58 [-3.00 to -2.16] | -2.26 [-2.69 to -1.84] | -2.27 [-2.69 to -1.84] | -2.58 [-3.00 to -2.16]
Statistical Analysis 1: Comparison: Standard Diet Monitoring vs Simplified Diet Monitoring; ITT analysis for factor 1 (dietary self-monitoring) using linear mixed models comparing the effect of standard dietary monitoring to simplified dietary monitoring on weight change over time (from baseline to 3 months); Test type: Superiority; p = 0.43, Mixed Models Analysis; DF (2,622); Mean Difference (Net) = 0.24, 95% CI 2-sided [-0.36 to 0.84] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Weekly Adaptive Activity Goals vs Daily Adaptive Activity Goals; ITT analysis for factor 2 (adaptive activity goals) using linear mixed models comparing the effect of weekly adaptive activity goals versus daily adaptive activity goals on weight change over time (from baseline to 3 months); Test type: Superiority; p = 0.17, Mixed Models Analysis; DF (2,622); Mean Difference (Net) = -0.42, 95% CI 2-sided [-1.01 to 0.18] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Fixed Message Decision Points vs Adaptive Message Decision Points; ITT analysis for factor 3 (message decision points) using linear mixed models comparing the effect of weekly adaptive activity goals versus daily adaptive activity goals on weight change over time (from baseline to 3 months); Test type: Superiority; p = 0.08, Mixed Models Analysis; DF (2,622); Mean Difference (Net) = 0.53, 95% CI 2-sided [-0.06 to 1.13] — [estimate comment as in outcome 1, analysis 3]
Statistical Analysis 4: Comparison: Standard Message Decision Rules vs Adaptive Message Decision Rules; ITT analysis for factor 4 (message decision rules) using linear mixed models comparing the effect of standard decision rules to adaptive decision rules on weight change over time (from baseline to 3 months); Test type: Superiority; p = 0.58, Mixed Models Analysis; DF (2,622); Mean Difference (Net) = 0.32, 95% CI 2-sided [-0.28 to 0.91] — [estimate comment as in outcome 1, analysis 4]
Statistical Analysis 5: Comparison: No Message Choice vs Message Choice; ITT analysis for factor 5 (participant choice) using linear mixed models comparing the effect of no participant message choice versus participant message choice on weight change over time (from baseline to 3 months); Test type: Superiority; p = 0.55, Mixed Models Analysis; DF (2,622); Mean Difference (Net) = -0.32, 95% CI 2-sided [-0.91 to 0.28] — [estimate comment as in outcome 1, analysis 5]

3. Secondary Outcome: Percent of Participants Reaching >/= 5% Weight Loss
Description: Percent change in body weight will be calculated (6 month weight - baseline weight/100) and determined to be at or above 5% indicating a clinically significant change.
Time Frame: Baseline to 6 months
Population: Participants with a 6-month weight value (total N = 583).
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Diet Monitoring | Simplified Diet Monitoring | Weekly Adaptive Activity Goals | Daily Adaptive Activity Goals | Fixed Message Decision Points | Adaptive Message Decision Points | Standard Message Decision Rules | Adaptive Message Decision Rules | No Message Choice | Message Choice
Number analyzed (Participants) | 289 | 294 | 294 | 289 | 295 | 288 | 294 | 289 | 293 | 290
Participants | 100 | 101 | 89 | 112 | 107 | 94 | 101 | 100 | 95 | 106
Statistical Analysis 1: Comparison: Standard Diet Monitoring vs Simplified Diet Monitoring; Chi-square test of the difference in proportion reaching 5% weight loss from baseline to 6 months between standard dietary monitoring and simplified dietary monitoring (factor 1); Test type: Superiority; p = 0.95, Chi-squared; DF (1); Odds Ratio (OR) = 0.99, 95% CI 2-sided [0.70 to 1.39] — Standard dietary monitoring coded as 0 (reference) and simplified dietary monitoring coded as 1; an odds ratio > 1 indicates that the odds of achieving 5% weight loss are higher in the group coded as 1
Statistical Analysis 2: Comparison: Weekly Adaptive Activity Goals vs Daily Adaptive Activity Goals; Chi-square test of the difference in proportion reaching 5% weight loss from baseline to 6 months between weekly adaptive activity goals and daily adaptive activity goals (factor 2); Test type: Superiority; p = 0.03, Chi-squared; DF (1); Odds Ratio (OR) = 1.46, 95% CI 2-sided [1.03 to 2.05] — Weekly adaptive activity goals coded as 0 (reference) and daily adaptive activity goals coded as 1; an odds ratio > 1 indicates that the odds of achieving 5% weight loss are higher in the group coded as 1
Statistical Analysis 3: Comparison: Fixed Message Decision Points vs Adaptive Message Decision Points; Chi-square test of the difference in proportion reaching 5% weight loss from baseline to 6 months between fixed message decision points and adaptive message decision points (factor 3); Test type: Superiority; p = 0.36, Chi-squared; DF (1); Odds Ratio (OR) = 0.85, 95% CI 2-sided [0.60 to 1.20] — Fixed decision points coded as 0 (reference) and adaptive decision points coded as 1; an odds ratio > 1 indicates that the odds of achieving 5% weight loss are higher in the group coded as 1
Statistical Analysis 4: Comparison: Standard Message Decision Rules vs Adaptive Message Decision Rules; Chi-square test of the difference in proportion reaching 5% weight loss from baseline to 6 months between standard message decision rules and adaptive message decision rules (factor 4); Test type: Superiority; p = 0.95, Chi-squared; DF (1); Odds Ratio (OR) = 1.01, 95% CI 2-sided [0.72 to 1.42] — Standard decision rules coded as 0 (reference) and adaptive decision rules coded as 1; an odds ratio > 1 indicates that the odds of achieving 5% weight loss are higher in the group coded as 1
Statistical Analysis 5: Comparison: No Message Choice vs Message Choice; Chi-square test of the difference in proportion reaching 5% weight loss from baseline to 6 months between no message choice and message choice (factor 5); Test type: Superiority; p = 0.29, Chi-squared; DF (1); Odds Ratio (OR) = 1.20, 95% CI 2-sided [0.85 to 1.69] — No message choice coded as 0 (reference) and message choice coded as 1; an odds ratio > 1 indicates that the odds of achieving 5% weight loss are higher in the group coded as 1

4. Secondary Outcome: Diet
Description: Change in daily caloric intake from baseline to 6 months as measured using the self-administered National Cancer Institute's Automated Self- Administered 24-hour Recall (ASA-24), a 24-hour recall that is self-administered on a week day and a weekend day at each timepoint. Change calculated as (daily kcal at 6 months - daily kcal at baseline).
Time Frame: Baseline, 6 months
Population: Participants who completed at least one 24-hour recall at 6 months (total N = 565).
Measure: Mean (Standard Deviation); unit: kcal/day
Arm/Group | Standard Diet Monitoring | Simplified Diet Monitoring | Weekly Adaptive Activity Goals | Daily Adaptive Activity Goals | Fixed Message Decision Points | Adaptive Message Decision Points | Standard Message Decision Rules | Adaptive Message Decision Rules | No Message Choice | Message Choice
Number analyzed (Participants) | 282 | 283 | 289 | 276 | 283 | 282 | 278 | 287 | 284 | 281
kcal/day | -378.6 (765.8) | -485.3 (813.4) | -470.3 (811.3) | -391.9 (768.8) | -452.3 (807.2) | -411.6 (775.5) | -439.7 (775.7) | -424.6 (807.1) | -476.9 (841.6) | -386.7 (735.3)

5. Secondary Outcome: Physical Activity
Description: Change in physical activity from baseline to 3 and 6 months as measured using the Paffenbarger Physical Activity Questionnaire (PPAQ). The PPAQ assesses amount of planned and lifestyle associated physical activity performed during a typical week. The PPAQ consists of three components: (1) stair climbing, (2) walking, and (3) sports and recreation. Participants report the frequency and duration of physical activity in the past week. Scoring yields energy expenditure from physical activity per week (kcal/week). Higher scores translate into greater energy expenditure per week (i.e.,better outcome). Range is 0 - no theoretical maximum. Outcome is change in kcal burned per week.
Time Frame: Baseline,3 months, 6 months
Population: Participants who completed the PPAQ at 3 months; participants who completed the PPAQ at 6 months.
Measure: Mean (Standard Deviation); unit: kcal/week
Arm/Group | Standard Diet Monitoring | Simplified Diet Monitoring | Weekly Adaptive Activity Goals | Daily Adaptive Activity Goals | Fixed Message Decision Points | Adaptive Message Decision Points | Standard Message Decision Rules | Adaptive Message Decision Rules | No Message Choice | Message Choice
Number analyzed (Participants) | 309 | 315 | 313 | 311 | 314 | 310 | 312 | 312 | 314 | 310
kcal/week
  Baseline to 3 Months: number analyzed (Participants) | 295 | 295 | 302 | 288 | 297 | 293 | 297 | 293 | 295 | 295
  Baseline to 3 Months | 180.4 (939.5) | 322.6 (1089.8) | 252.1 (967.1) | 250.8 (1072.5) | 309.3 (1074.4) | 192.9 (957.8) | 268.0 (1075.3) | 234.8 (960.1) | 149.8 (934.7) | 353.2 (1089.0)
  Baseline to 6 Months: number analyzed (Participants) | 283 | 285 | 289 | 279 | 288 | 280 | 283 | 285 | 287 | 281
  Baseline to 6 Months | 167.1 (927.9) | 92.1 (861.5) | 128.0 (899.1) | 131.0 (892.7) | 163.6 (911.8) | 94.4 (878.0) | 131.7 (899.5) | 127.3 (892.4) | 102.9 (854.0) | 156.6 (936.2)

6. Secondary Outcome: Sedentary Behavior Score
Description: Change in sedentary behavior from baseline to 3 and 6 months as measured using the 12- item Sedentary Behavior Questionnaire which asks respondents to indicate the number of hours they spend on a typical weekday and a typical weekend day doing each of six activities. The scale ranges from "none" to "6 or more hours" for each item. Higher values on the Sedentary Behavior Questionnaire indicate greater amount of time spent in sedentary behavior. Range is 0 to 24 hours and outcome is change in minutes per day.
Time Frame: Baseline, 3 months, 6 months
Population: Participants who completed the Sedentary Behavior Questionnaire at 3 months; participants who completed the Sedentary Behavior Questionnaire at 6 months.
Measure: Mean (Standard Deviation); unit: minutes/day
Arm/Group | Standard Diet Monitoring | Simplified Diet Monitoring | Weekly Adaptive Activity Goals | Daily Adaptive Activity Goals | Fixed Message Decision Points | Adaptive Message Decision Points | Standard Message Decision Rules | Adaptive Message Decision Rules | No Message Choice | Message Choice
Number analyzed (Participants) | 309 | 315 | 313 | 311 | 314 | 310 | 312 | 312 | 314 | 310
minutes/day
  Baseline to 3 Months: number analyzed (Participants) | 292 | 295 | 300 | 287 | 295 | 292 | 295 | 292 | 295 | 292
  Baseline to 3 Months | -35.3 (207.6) | -36.1 (223.4) | -33.9 (194.0) | -37.6 (236.2) | -41.1 (200.9) | -30.3 (229.5) | -40.9 (217.3) | -30.5 (213.9) | -34.1 (222.9) | -37.4 (208.1)
  Baseline to 6 Months: number analyzed (Participants) | 283 | 285 | 289 | 279 | 288 | 280 | 283 | 285 | 287 | 281
  Baseline to 6 Months | -22.7 (218.9) | -34.1 (227.0) | -11.8 (223.7) | -45.7 (221.1) | -39.9 (223.7) | -16.6 (221.8) | -28.3 (230.1) | -28.6 (215.9) | -28.3 (236.8) | -28.5 (208.1)

7. Secondary Outcome: Autonomy Support Score
Description: Autonomy support at 3 and 6 months. Items are adapted from the Health Care Climate Questionnaire, which is a measure of how the participant perceives support from a healthcare provider, to measure autonomy support from the program. The scale includes 15 items rated on a scale of 1 (strongly disagree) to 7 (strongly agree) (e.g., "I feel that [the program] has provided me choices and options.") Scores are calculated by averaging the individual item scores (with item 13 reverse-scored). Higher average scores represent a higher level of perceived autonomy support. Outcomes are the mean value at 3 months and the mean value at 6 months.
Time Frame: 3 months, 6 months
Population: Participants who completed the Health Care Climate Questionnaire at 3 months; participants who completed the Health Care Climate Questionnaire at 6 months.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Diet Monitoring | Simplified Diet Monitoring | Weekly Adaptive Activity Goals | Daily Adaptive Activity Goals | Fixed Message Decision Points | Adaptive Message Decision Points | Standard Message Decision Rules | Adaptive Message Decision Rules | No Message Choice | Message Choice
Number analyzed (Participants) | 309 | 315 | 313 | 311 | 314 | 310 | 312 | 312 | 314 | 310
score on a scale
  3 Months: number analyzed (Participants) | 293 | 294 | 299 | 288 | 295 | 292 | 295 | 292 | 295 | 292
  3 Months | 5.14 (1.20) | 5.11 (1.11) | 5.08 (1.15) | 5.17 (1.15) | 5.16 (1.15) | 5.09 (1.16) | 5.12 (1.17) | 5.13 (1.13) | 5.13 (1.15) | 5.12 (1.15)
  6 Months: number analyzed (Participants) | 284 | 285 | 284 | 278 | 287 | 286 | 280 | 279 | 281 | 281
  6 Months | 5.13 (1.22) | 5.08 (1.30) | 5.05 (1.25) | 5.12 (1.28) | 5.08 (1.23) | 5.11 (1.26) | 5.12 (1.22) | 5.09 (1.25) | 5.07 (1.29) | 5.15 (1.26)

8. Secondary Outcome: Competence for Diet and Physical Activity Scores
Description: Change in perceived competence from baseline to 3 and 6 months as measured using the The Perceived Competence Scale. The Scale measures perceived competence for diet (4 items) and physical activity (4 items). Items are rated on a 7-point Likert scale (1 = not at all true, 7 = very true), and include items such as "I feel confident in my ability to maintain a healthy diet." Scores are summed for the items in the subscale (diet and physical activity) and the range for each subscale is 4 - 28. Greater values indicate higher levels of perceived competence for engaging in positive diet and physical activity behaviors. Scores are summed for the items in each subscale separately (diet and physical activity). Outcomes are change in perceived competence for diet and change in perceived competence for physical activity.
Time Frame: Baseline, 3 months, 6 months
Population: Participants who completed the Perceived Competence Scale for Diet at 3 months; participants who completed the Perceived Competence Scale for Diet at 6 months.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Diet Monitoring | Simplified Diet Monitoring | Weekly Adaptive Activity Goals | Daily Adaptive Activity Goals | Fixed Message Decision Points | Adaptive Message Decision Points | Standard Message Decision Rules | Adaptive Message Decision Rules | No Message Choice | Message Choice
Number analyzed (Participants) | 309 | 315 | 313 | 311 | 314 | 310 | 312 | 312 | 314 | 310
score on a scale
  Competence for Diet - Baseline to 3 Months: number analyzed (Participants) | 293 | 295 | 301 | 287 | 296 | 292 | 296 | 292 | 295 | 293
  Competence for Diet - Baseline to 3 Months | 0.88 (6.01) | 0.74 (6.36) | 0.41 (6.17) | 1.23 (6.17) | 0.78 (6.22) | 0.84 (6.15) | 1.32 (5.66) | 0.29 (6.64) | 0.62 (6.05) | 1.00 (6.32)
  Competence for Diet - Baseline to 6 Months: number analyzed (Participants) | 283 | 284 | 288 | 279 | 287 | 280 | 283 | 284 | 287 | 280
  Competence for Diet - Baseline to 6 Months | 2.03 (6.76) | 1.62 (6.81) | 1.74 (6.75) | 1.90 (6.83) | 1.91 (6.97) | 1.74 (6.60) | 2.26 (6.51) | 1.38 (7.03) | 1.81 (6.83) | 1.83 (6.75)
  Competence for Physical Activity - Baseline to 3 Months: number analyzed (Participants) | 293 | 295 | 301 | 287 | 296 | 292 | 296 | 292 | 295 | 293
  Competence for Physical Activity - Baseline to 3 Months | -0.83 (6.51) | -1.50 (6.09) | -1.10 (6.37) | -1.23 (6.25) | -1.27 (6.36) | -1.06 (6.26) | -0.92 (6.28) | -1.42 (6.33) | -1.02 (6.55) | -1.31 (6.05)
  Competence for Physical Activity - Baseline to 6 Months: number analyzed (Participants) | 283 | 284 | 288 | 279 | 287 | 280 | 283 | 284 | 287 | 280
  Competence for Physical Activity - Baseline to 6 Months | -0.14 (6.67) | -1.18 (6.57) | -0.87 (6.65) | -0.44 (6.62) | -0.87 (6.84) | -0.45 (6.41) | -0.40 (6.40) | -0.92 (6.86) | -0.31 (7.03) | -1.03 (6.20)

9. Secondary Outcome: Perceived Message Relevance Score
Description: Perceived message relevance at 3 and 6 months as measured using two items used in our previous work and adapted from previous studies of tailored messages. Participants were asked to rate how strongly they disagree or agree with the statements about messages being "written personally for me" and "applied to my life." Responses are on a 5-point scale from 1 (strongly disagree) to 5 (strongly agree). The values of the two items are averaged for a final score. Higher values indicate that a participant perceives the messages received in the program are more relevant to them.
Time Frame: 3 months, 6 months
Population: Participants who completed message relevance items at 3 months; participants who completed message relevance items at 6 months.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Diet Monitoring | Simplified Diet Monitoring | Weekly Adaptive Activity Goals | Daily Adaptive Activity Goals | Fixed Message Decision Points | Adaptive Message Decision Points | Standard Message Decision Rules | Adaptive Message Decision Rules | No Message Choice | Message Choice
Number analyzed (Participants) | 309 | 315 | 313 | 311 | 314 | 310 | 312 | 312 | 314 | 310
score on a scale
  3 Months: number analyzed (Participants) | 293 | 294 | 299 | 288 | 295 | 292 | 295 | 292 | 295 | 292
  3 Months | 3.34 (0.97) | 3.37 (0.95) | 3.29 (0.94) | 3.42 (0.98) | 3.35 (0.98) | 3.36 (0.94) | 3.35 (0.96) | 3.36 (0.96) | 3.40 (0.96) | 3.31 (0.96)
  6 Months: number analyzed (Participants) | 281 | 284 | 287 | 278 | 285 | 280 | 281 | 284 | 286 | 279
  6 Months | 3.36 (1.01) | 3.33 (1.05) | 3.35 (0.99) | 3.35 (1.07) | 3.37 (1.01) | 3.33 (1.05) | 3.34 (1.04) | 3.36 (1.02) | 3.36 (1.05) | 3.33 (1.01)

10. Secondary Outcome: Treatment Self-Regulation Score
Description: Change in treatment self-regulation from baseline to 3 and 6 months as measured using the Treatment Self-Regulation Questionnaire (TSRQ). The TSRQ assesses autonomous and controlled motivation for making changes in diet (15 items) and physical activity (15 items). Examples item: "Because I feel that I want to take responsibility for my own health" answered on a scale of 1 (not at all true) to 7 (very true)." Calculating the scores for the sub-scales will consist of averaging the items on that subscale. They are:
  Autonomous Regulation: 2, 3, 7, 10, 13, 16, 18, 19 Controlled Regulation: 1, 4, 5, 6, 8, 9, 11, 12, 14, 15, 17. Responses to the items within the subscale are averaged with the range of scores being 1 to 7. Higher values on each subscale indicate greater levels of that type of motivation. Outcomes are changes in autonomous and controlled motivation for diet at 3 and 6 months, and changes in autonomous and controlled motivation for activity at 3 and 6 months.
Time Frame: Baseline, 3 months, 6 months
Population: Participants who completed the TSRQ at 3 months; participants who completed the TSRQ at 6 months.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Diet Monitoring | Simplified Diet Monitoring | Weekly Adaptive Activity Goals | Daily Adaptive Activity Goals | Fixed Message Decision Points | Adaptive Message Decision Points | Standard Message Decision Rules | Adaptive Message Decision Rules | No Message Choice | Message Choice
Number analyzed (Participants) | 309 | 315 | 313 | 311 | 314 | 310 | 312 | 312 | 314 | 310
score on a scale
  Autonomous motivation for diet baseline to 3 months: number analyzed (Participants) | 292 | 294 | 299 | 287 | 295 | 291 | 295 | 291 | 294 | 292
  Autonomous motivation for diet baseline to 3 months | -0.19 (0.93) | -0.23 (0.87) | -0.16 (0.87) | -0.25 (0.92) | -0.19 (0.85) | -0.22 (0.94) | -0.21 (0.90) | -0.20 (0.90) | -0.18 (0.89) | -0.23 (0.91)
  Autonomous motivation for diet baseline to 6 months: number analyzed (Participants) | 281 | 284 | 287 | 278 | 285 | 280 | 281 | 284 | 286 | 279
  Autonomous motivation for diet baseline to 6 months | -0.17 (1.06) | -0.18 (0.98) | -0.12 (0.97) | -0.23 (1.07) | -0.14 (1.00) | -0.21 (1.05) | -0.20 (1.08) | -0.15 (0.97) | -0.17 (1.02) | -0.18 (1.03)
  Controlled motivation for diet baseline to 3 months: number analyzed (Participants) | 292 | 294 | 299 | 287 | 295 | 291 | 295 | 291 | 294 | 292
  Controlled motivation for diet baseline to 3 months | 0.16 (1.10) | 0.06 (1.20) | 0.15 (1.17) | 0.06 (1.13) | 0.07 (1.15) | 0.14 (1.15) | 0.09 (1.06) | 0.13 (1.24) | 0.02 (1.17) | 0.20 (1.12)
  Controlled motivation for diet baseline to 6 months: number analyzed (Participants) | 281 | 284 | 287 | 278 | 285 | 280 | 281 | 284 | 286 | 279
  Controlled motivation for diet baseline to 6 months | 0.17 (1.17) | 0.07 (1.16) | 0.16 (1.16) | 0.08 (1.17) | 0.12 (1.16) | 0.12 (1.17) | 0.17 (1.11) | 0.07 (1.22) | 0.03 (1.15) | 0.21 (1.17)
  Autonomous motivation for physical activity baseline to 3 months: number analyzed (Participants) | 294 | 295 | 301 | 288 | 296 | 293 | 297 | 292 | 295 | 294
  Autonomous motivation for physical activity baseline to 3 months | -0.07 (1.04) | -0.06 (0.94) | -0.07 (0.94) | -0.06 (1.04) | -0.02 (0.96) | -0.11 (1.02) | -0.02 (0.99) | -0.12 (0.99) | -0.03 (0.97) | -0.10 (1.01)
  Autonomous motivation for physical activity baseline to 6 months: number analyzed (Participants) | 283 | 284 | 288 | 279 | 287 | 280 | 283 | 284 | 287 | 280
  Autonomous motivation for physical activity baseline to 6 months | -0.01 (1.07) | 0.03 (1.02) | 0.01 (0.91) | 0.02 (1.17) | 0.08 (1.00) | -0.06 (1.09) | 0.00 (1.12) | 0.03 (0.97) | 0.04 (1.09) | -0.02 (1.00)
  Controlled motivation for physical activity baseline to 3 months: number analyzed (Participants) | 294 | 295 | 301 | 288 | 296 | 293 | 297 | 292 | 295 | 294
  Controlled motivation for physical activity baseline to 3 months | 0.07 (1.14) | 0.14 (1.03) | 0.17 (1.04) | 0.04 (1.13) | 0.09 (1.03) | 0.12 (1.14) | 0.06 (1.03) | 0.16 (1.14) | 0.08 (1.08) | 0.13 (1.09)
  Controlled motivation for physical activity baseline to 6 months: number analyzed (Participants) | 283 | 284 | 288 | 279 | 287 | 280 | 283 | 284 | 287 | 280
  Controlled motivation for physical activity baseline to 6 months | 0.06 (1.11) | 0.17 (1.11) | 0.15 (1.10) | 0.08 (1.13) | 0.16 (1.07) | 0.07 (1.15) | 0.10 (1.08) | 0.14 (1.14) | 0.06 (1.10) | 0.17 (1.12)

11. Secondary Outcome: Relatedness Score
Description: Relatedness at 3 and 6 months as measured with 3 items adapted from the 8-item Relatedness subscale of the Basic Need Satisfaction at Work Scale. Examples include "The messages demonstrate caring about me as a person" and are scored on a Likert scale from 1 (strongly disagree) to 7 (strongly agree). Responses are averaged with a range of 1 to 7. Higher scores indicate a higher level of perceived relatedness from the intervention messages.
Time Frame: 3 months, 6 months
Population: Participants who completed the relatedness subscale at 3 months; participants who completed the relatedness subscale at 6 months.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Diet Monitoring | Simplified Diet Monitoring | Weekly Adaptive Activity Goals | Daily Adaptive Activity Goals | Fixed Message Decision Points | Adaptive Message Decision Points | Standard Message Decision Rules | Adaptive Message Decision Rules | No Message Choice | Message Choice
Number analyzed (Participants) | 309 | 315 | 313 | 311 | 314 | 310 | 312 | 312 | 314 | 310
score on a scale
  Relatedness at 3 Months: number analyzed (Participants) | 293 | 294 | 299 | 288 | 295 | 292 | 295 | 292 | 295 | 292
  Relatedness at 3 Months | 4.91 (1.47) | 4.95 (1.40) | 4.86 (1.42) | 5.01 (1.45) | 4.99 (1.42) | 4.88 (1.45) | 4.91 (1.40) | 4.96 (1.48) | 5.04 (1.43) | 4.83 (1.44)
  Relatedness at 6 Months: number analyzed (Participants) | 281 | 284 | 287 | 278 | 285 | 280 | 281 | 284 | 286 | 279
  Relatedness at 6 Months | 4.79 (1.57) | 4.90 (1.51) | 4.83 (1.50) | 4.85 (1.58) | 4.91 (1.52) | 4.77 (1.56) | 4.86 (1.53) | 4.83 (1.55) | 4.93 (1.52) | 4.75 (1.55)

12. Secondary Outcome: Diet Self-monitoring Adherence
Description: Mean number of days of complete dietary tracking summed over the 6-month study period.
Time Frame: Baseline to 6 months (daily)
Population: All randomized participants.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Standard Diet Monitoring | Simplified Diet Monitoring | Weekly Adaptive Activity Goals | Daily Adaptive Activity Goals | Fixed Message Decision Points | Adaptive Message Decision Points | Standard Message Decision Rules | Adaptive Message Decision Rules | No Message Choice | Message Choice
Number analyzed (Participants) | 309 | 315 | 313 | 311 | 314 | 310 | 312 | 312 | 314 | 310
days | 73.3 (51.3) | 67.9 (48.1) | 69.3 (50.1) | 71.9 (49.4) | 69.2 (49.1) | 72.1 (50.4) | 74.9 (51.4) | 66.3 (47.6) | 69.7 (50.4) | 71.5 (49.0)

13. Secondary Outcome: Weighing Adherence
Description: Mean number of days of self-weighing over the 6 month period.
Time Frame: Baseline to 6 months (daily)
Population: All randomized participants.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Standard Diet Monitoring | Simplified Diet Monitoring | Weekly Adaptive Activity Goals | Daily Adaptive Activity Goals | Fixed Message Decision Points | Adaptive Message Decision Points | Standard Message Decision Rules | Adaptive Message Decision Rules | No Message Choice | Message Choice
Number analyzed (Participants) | 309 | 315 | 313 | 311 | 314 | 310 | 312 | 312 | 314 | 310
days | 90.2 (51.4) | 87.4 (49.6) | 87.5 (50.9) | 90.0 (50.1) | 87.9 (50.6) | 89.6 (50.5) | 90.5 (51.2) | 87.0 (49.8) | 88.6 (50.8) | 89.0 (50.3)

14. Secondary Outcome: Physical Activity Self-monitoring Adherence
Description: Mean number of days of physical activity tracking over the 6 month period as measured by Fitbit tracker wear.
Time Frame: Baseline to 6 months (daily)
Population: All randomized participants.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Standard Diet Monitoring | Simplified Diet Monitoring | Weekly Adaptive Activity Goals | Daily Adaptive Activity Goals | Fixed Message Decision Points | Adaptive Message Decision Points | Standard Message Decision Rules | Adaptive Message Decision Rules | No Message Choice | Message Choice
Number analyzed (Participants) | 309 | 315 | 313 | 311 | 314 | 310 | 312 | 312 | 314 | 310
days | 134.1 (46.5) | 133.4 (45.3) | 133.2 (46.3) | 134.3 (45.4) | 132.7 (46.7) | 134.8 (45.0) | 133.9 (45.9) | 133.6 (45.8) | 131.4 (48.2) | 136.2 (43.2)

ADVERSE EVENTS:
Time Frame: up to 6 months
Arm/Group | Condition 1 | Condition 2 | Condition 3 | Condition 4 | Condition 5 | Condition 6 | Condition 7 | Condition 8 | Condition 9 | Condition 10 | Condition 11 | Condition 12 | Condition 13 | Condition 14 | Condition 15 | Condition 16 | Condition 17 | Condition 18 | Condition 19 | Condition 20 | Condition 21 | Condition 22 | Condition 23 | Condition 24 | Condition 25 | Condition 26 | Condition 27 | Condition 28 | Condition 29 | Condition 30 | Condition 31 | Condition 32
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/21 | 0/20 | 0/18 | 0/20 | 0/18 | 0/19 | 0/20 | 0/20 | 0/20 | 1/20 | 2/19 | 0/18 | 1/19 | 0/20 | 0/19 | 0/20 | 0/20 | 0/20 | 2/19 | 0/20 | 1/19 | 0/20 | 0/19 | 1/19 | 1/20 | 0/20 | 0/20 | 0/20 | 0/20 | 0/20 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/21 | 0/20 | 0/18 | 0/20 | 0/18 | 0/19 | 0/20 | 1/20 | 0/20 | 1/20 | 1/19 | 0/18 | 1/19 | 0/20 | 0/19 | 0/20 | 0/20 | 0/20 | 2/19 | 0/20 | 1/19 | 0/20 | 0/19 | 1/19 | 1/20 | 0/20 | 0/20 | 0/20 | 0/20 | 0/20 | 0/19
Other Adverse Events (participants affected / at risk) | 5/18 | 2/21 | 3/20 | 5/18 | 2/20 | 4/18 | 1/19 | 3/20 | 4/20 | 7/20 | 4/20 | 1/19 | 2/18 | 3/19 | 2/20 | 4/19 | 3/20 | 1/20 | 1/20 | 3/19 | 2/20 | 4/19 | 2/20 | 0/19 | 5/19 | 3/20 | 3/20 | 2/20 | 4/20 | 6/20 | 1/20 | 5/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Condition 1 (N=18) | Condition 2 (N=21) | Condition 3 (N=20) | Condition 4 (N=18) | Condition 5 (N=20) | Condition 6 (N=18) | Condition 7 (N=19) | Condition 8 (N=20) | Condition 9 (N=20) | Condition 10 (N=20) | Condition 11 (N=20) | Condition 12 (N=19) | Condition 13 (N=18) | Condition 14 (N=19) | Condition 15 (N=20) | Condition 16 (N=19) | Condition 17 (N=20) | Condition 18 (N=20) | Condition 19 (N=20) | Condition 20 (N=19) | Condition 21 (N=20) | Condition 22 (N=19) | Condition 23 (N=20) | Condition 24 (N=19) | Condition 25 (N=19) | Condition 26 (N=20) | Condition 27 (N=20) | Condition 28 (N=20) | Condition 29 (N=20) | Condition 30 (N=20) | Condition 31 (N=20) | Condition 32 (N=19)
Miscarriage (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — hospitalized overnight
Leg injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hospitalized for transient ischemic attacks (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gall bladder removal (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis, surgery and hospitalization (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Surgery (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — no other detail provided by participant
Ileostomy secondary to parastomal hernia (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — surgery and hospitalization
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Condition 1 (N=18) | Condition 2 (N=21) | Condition 3 (N=20) | Condition 4 (N=18) | Condition 5 (N=20) | Condition 6 (N=18) | Condition 7 (N=19) | Condition 8 (N=20) | Condition 9 (N=20) | Condition 10 (N=20) | Condition 11 (N=20) | Condition 12 (N=19) | Condition 13 (N=18) | Condition 14 (N=19) | Condition 15 (N=20) | Condition 16 (N=19) | Condition 17 (N=20) | Condition 18 (N=20) | Condition 19 (N=20) | Condition 20 (N=19) | Condition 21 (N=20) | Condition 22 (N=19) | Condition 23 (N=20) | Condition 24 (N=19) | Condition 25 (N=19) | Condition 26 (N=20) | Condition 27 (N=20) | Condition 28 (N=20) | Condition 29 (N=20) | Condition 30 (N=20) | Condition 31 (N=20) | Condition 32 (N=19)
Palpitations from anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ankle sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthma attacks/exacerbation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back sprain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
ADHD (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fainting (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Foot pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Knee sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nerve inflammation, wrist and hand (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Heart palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
High blood pressure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intracranial Hypertension and Neurogenic Thoracic Outlet Syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Knee injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Finger injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Miscarriage (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Motor vehicle accident (General disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hand and wrist pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neck and shoulder pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diabetes (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Heart trouble (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — no other details provided
Wrist sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deltoid sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Shin splints (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toe sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nerve pain/sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eating disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PTSD, started medication (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest muscle strain secondary to pneumonia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle strain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toe injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wisdom tooth removal (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
WPW syndrome (congenital heart defect) (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Breathing problems (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Due to motor vehicle accident
Switched medication for mental health disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sternum injury (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Other mental health treatment (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neck, back, and shoulder injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Due to motor vehicle accident

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-02-20): https://cdn.clinicaltrials.gov/large-docs/16/NCT04922216/Prot_SAP_001.pdf
  • Informed Consent Form (2023-02-20): https://cdn.clinicaltrials.gov/large-docs/16/NCT04922216/ICF_002.pdf